# **Prediction of Findings From the Ongoing PRONOUNCE Trial Using Healthcare Database Analyses**

# **DUPLICATE - PRONOUNCE**

September 9, 2021

NCT04897958

#### 1. RCT Details

This section provides a high-level overview of a **published** RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Cardiovascular Safety of Degarelix Versus Leuprolide for Advanced Prostate Cancer (PRONOUNCE Trial)

# 1.2 <u>Intended aim(s)</u>

To compare the incidence of major cardiovascular events (MACE) among advanced prostate cancer subjects treated with degarelix versus leuprolide.

# 1.3 Primary endpoint for replication

Time from randomization to the first confirmed, adjudicated occurrence of a MACE, which is defined as a composite of all-cause death, nonfatal myocardial infarction, or nonfatal stroke through 12 months of ADT treatment.

## 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

Based on prior literature, it was determined that 66 MACE events and 876 subjects would be required to reject a two-sided null hypothesis of equal hazards with 80% power at a 5% type I error rate. A hazard ratio of 0.49 with absolute event rates of 5.1% and 10.2% (degarelix vs leuprolide) were hypothesized.

# 1.5 Secondary endpoint for replication (assay sensitivity) and RCT finding

Secondary cardiovascular objectives: To assess 1) the frequency of MACE components individually (i.e., nonfatal myocardial infarction, nonfatal stroke, and all-cause mortality)

# 1.6 Trial estimate

The trial is ongoing and scheduled to complete in April 2021.

# 2. Person responsible for implementation of replication in Aetion

David Merola, PharmD, SM and Sushama Kattinakere Sreedhara, MBBS, MSPH, implemented the study design in the Aetion Evidence Platform. They are not responsible for the validity of the design and analytic choices. All implementation steps are recorded, and the implementation history is archived in the platform.

# 3. Data Source(s)

Optum CDM, IBM® MarketScan®, Medicare Diabetes

# 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Figure 1.



#### 5. Cohort Identification

#### 5.1 Cohort Summary

An active-comparator, incident-user design will be employed to compare patients that received degarelix vs. leuprolide. Subjects will be selected on the basis of having at least one diagnosis code indicating prostate cancer, male sex, and a history of atherosclerotic cardiovascular disease. Subjects will be excluded if they were not treatment-naïve with respect to prostate cancer, had a record of uncontrolled diabetes or hypertension within 30 days prior to treatment initiation, had a history of long QT syndrome or risk factors thereof (i.e., heart failure, hypokalemia, or medications known to prolong the QT interval), or an acute myocardial infarction, stroke, or revascularization procedure within 30 days prior to treatment initiation. In contrast to the PRONOUNCE trial, patients cannot be required to have had established tumor staging information, angiography-verified stenosis/occlusion of vessels, and a lack of planned cardiac surgery at the time of treatment initiation due to poor capture of this information in administrative data. All patients were required to have continuous enrollment for 365 days prior to cohort entry to ensure incident use of the study drugs.

#### 5.2 Important steps for cohort formation

Incident use of the exposure (leuprolide or degarelix) is defined as no use of the exposure drug in the 365 days prior to meeting all eligibility criteria and initiation of exposure.

# 5.2.1 Eligible cohort entry dates

The degarelix indication for treatment of prostate cancer was approved by the FDA on Dec 24, 2008. Leuprolide was initially approved for the same indication prior to Dec 24, 2008.

- IBM® MarketScan®: Dec 24, 2008 December 31, 2018 (end of available data)
- Optum CDM: Dec 24, 2008 June 30, 2020 (end of available data)
- CMS Diabetes: Dec 24, 2008 Dec 31, 2017 (end of available data)
- 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix** and are summarized in the flowcharts below.

# 5.3 Flowchart of the study cohort assembly

For Degarelix vs Leuprolide

| | IBM® Mar | ketScan® | Optum | CDM | CMS - D | iabetes |
|---|---|---|---|---|---|---|
| | Less Excluded Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients in our database | | 200,203,908 | | 78,202,636 | | 23,466,175 |
| Patients with Degarelix/Leuprolide [measured between Dec 24, 2008 and Dec 31, 2019.] | -199,937,514 | 266,394 | -78,046,787 | 155,849 | -23,212,628 | 253,547 |
| Excluded due to insufficient enrollment [-365, 0] | -94,870 | 171,524 | -36,242 | 119,607 | -125,589 | 127,958 |
| After wash-out for prior use of reference (Leuprolide) [-365, -1] | -106,281 | 65,243 | -77,869 | 41,738 | -96,813 | 31,145 |
| After wash-out for prior use of exposure (Degarelix) [-365, -1] and Excluded because patient qualified in >1 exposure category | -1,961 | 63,282 | -2,153 | 39,585 | -3,397 | 27,748 |
| Inclusion only Male gender [-365, 0] | -43,683 | 19,599 | -17,401 | 22,184 | -183 | 27,565 |
| <b>Inclusion Prostate Cancer</b> [start of all available data, 0] | -784 | 18,815 | -502 | 21,682 | -210 | 27,355 |
| Inclusion Pre-existing ASCVD [start of all available data, -30] | -14,187 | 4,628 | -15,729 | 5,953 | -16,099 | 11,256 |
| Exclusion Androgen deprivation therapy (GnRH agonists/antagonists) [-365, 0] | -145 | 4,483 | -106 | 5,847 | -465 | 10,791 |
| Exclusion Androgen deprivation therapy (hormonal therapy) [-365, -14] and Exclusion Androgen deprivation therapy (Orchiectomy) [start of all available data, 0] | -575 | 3,908 | -748 | 5,099 | -1,768 | 9,023 |
| Exclusion Uncontrolled Diabetes [-30, 0] | 0 | 3,908 | 0 | 5,099 | 0 | 9,023 |
| Exclusion Uncontrolled Hypertension [-30, 0] | -28 | 3,880 | -19 | 5,080 | -97 | 8,926 |
| <b>Exclusion Heart failure</b> [starts of all available data, 0] | -285 | 3,595 | -556 | 4,524 | -1,602 | 7,324 |
| <b>Exclusion QT syndrome</b> [starts of all available data, 0] | -7 | 3,588 | -9 | 4,515 | -19 | 7,305 |

| Exclusion Hypokalemia [-90, 0] | -3 | 3,585 | -14 | 4,501 | -37 | 7,268 |
|---|---|---|---|---|---|---|
| Exclusion Hypomagnesemia [-90, 0] | -9 | 3,576 | -7 | 4,494 | -12 | 7,256 |
| Exclusion QT prolonging medicines [0, 0] | -192 | 3,384 | -191 | 4,303 | -446 | 6,810 |
| Exclusion Acute MI [-29, 0] | -6 | 3,378 | -9 | 4,294 | -11 | 6,799 |
| Exclusion Stroke [-29, 0] and Exclusion Revascularization [-29,0] | -9 | 3,369 | -16 | 4,278 | -29 | 6,770 |
| Final cohort | | 3,369 | | 4,278 | | 6,770 |

<sup>\*\*</sup>Certain exclusion criteria are in collapsed form to maintain compliance with CMS' cell suppression policy\*\*

#### 6. Variables

#### 6.1 Exposure-related variables:

#### Study drug:

The study exposure of interest is defined by a HCPCS/CPT code or outpatient prescription drug claim indicating degarelix administration or dispensation, respectively. New initiation will be defined by no such records of degarelix in the prior 365 days before treatment initiation (washout period) and fulfillment of study eligibility criteria.

## **Comparator agent:**

The comparator is defined by an HCPCS/CPT code or outpatient prescription drug claim indicating leuprolide administration or dispensation, respectively. New initiation will be defined by no such records of leuprolide in the prior 365 days before treatment initiation (washout period) and fulfillment of study eligibility criteria.

# 6.2 Preliminary Covariates:

#### Age

The covariate listed above represents only a small subset of the covariate vector that will ultimately be controlled for in the design and analysis. We use the covariate above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (**Appendix B**). Gender is not included since the study is already restricted to male subjects.

#### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcome variables of interest (definitions provided in **Appendix**):

- **Primary outcome:** MACE (all-cause death, nonfatal myocardial infarction, or nonfatal stroke through 12 months of primary treatment with leuprolide or degarelix)
- Secondary outcomes:
  - Secondary cardiovascular objectives: To assess 1) the frequency of MACE components individually (i.e., nonfatal myocardial infarction, nonfatal stroke, and all-cause mortality)

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on day of cohort entry. An allowable gap of 90 days between records indicating each treatment will qualify as "continuous therapy" with respect to follow-up in the as-treated analysis.

The follow-up will start the day after drug initiation (i.e., cohort entry date), and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- 365 days
- Switch
- Discontinuation (90 days allowable grace period and risk window)

In the secondary ITT analysis, we will not censor for discontinuation or switching among study drugs

# 7. Initial Feasibility Analysis

## Aetion report name:

For degarelix vs. leuprolide

Optum CDM- https://bwh-dope.aetion.com/projects/details/1636/rwrs/67085

IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1323/rwrs/67083

CMS Diabetes - https://bwh-dope.aetion.com/projects/details/1637/rwrs/67081

Date conducted: 03/06/2021

Complete Aetion feasibility analysis using age as the only covariate and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed, nor will incidence rates be stratified by treatment group.

• Report patient characteristics by treatment group

Degarelix vs Leuprolide

| | C | Optum CDM | | IBM® MarketScan® | | CMS - Diabetes | | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Leuprolide -<br>Comparator | Degarelix -<br>Exposure | Difference | Leuprolide -<br>Comparator | Degarelix -<br>Exposure | Difference | Leuprolide -<br>Comparator | Degarelix -<br>Exposure | Difference |
| Number of patients | 3,676 | 596 | | 2,936 | 431 | | 5,828 | 941 | |
| Age | | | | | | | | | |
| mean<br>(sd) | 75.71 (7.42) | 75.93 (7.66) | -0.22 (-0.88,<br>0.44) | 74.38 (9.05) | 74.49 (9.12) | -0.11 (-1.03,<br>0.82) | 76.85 (6.58) | 76.94 (6.49) | -0.09 (-0.53,<br>0.36) |
| median<br>[IQR] | 76.00 [71.00,<br>81.00] | 76.00<br>[71.00,<br>82.00] | | 75.00 [68.00,<br>81.00] | 75.00<br>[68.00,<br>82.00] | | 76.00 [72.00,<br>81.00] | 77.00<br>[72.00,<br>81.87] | |

- Report summary parameters of study population FEASIBILITY- FOR STUDY OUTCOME
  - For Degarelix vs Leuprolide

| FEASIBILITY FOR STUDY OUTCOME | | | |
|---|---|---|---|
| | Optum CDM | IBM® MarketScan® | CMS - Diabetes |
| Number of patients in full cohort | 4,278 | 3,369 | 6,770 |
| Number of patients dropped as incomplete cases | 0 | 0 | 0 |
| Number of patients that did not begin follow-up | 6 | 2 | 1 |
| Number of patients in analytic cohort | 4,272 | 3,367 | 6,769 |
| Number of events | 108 | 43 | 211 |
| Number of person-years | 1,259.68 | 1,001.03 | 2,031.94 |
| Number of patients in group: Leuprolide - Comparator | 3,676 | 2,936 | 5,828 |
| Number of patients in group: Degarelix - Exposure | 596 | 431 | 941 |
| Risk per 1,000 patients | 25.28 | 12.77 | 31.17 |
| Rate per 1,000 person-years | 85.74 | 42.96 | 103.84 |

- Report median follow-up time by treatment group
  - For Degarelix vs Leuprolide

| FOLLOW-UP TIME FOR STUDY OUTCOME Median Follow-Up Time (Days) [IQR] – At 90 days gap | | | |
|---|---|---|---|
| Patient Group Optum CDM IBM® MarketScan® CMS - Diabetes | | | |
| Overall Patient Population | 89 [89, 89] | 89 [89, 89] | 89 [89, 89] |
| Referent - Leuprolide 89 [89, 89] 89 [89, 89] 89 [89, 89] | | | |
| Exposure - Degarelix | 82 [33, 132] | 68 [31, 126] | 67 [32, 124] |

- Report reasons for censoring in the overall study population
  - For Degarelix vs Leuprolide

| CENSORING REASONS FOR STUDY OUTCOME | | | |
|---|---|---|---|
| Reasons | Optum CDM | IBM® MarketScan® | CMS - Diabetes |
| Outcome | 108 (2.5%) | 43 (1.3%) | 211 (3.1%) |
| Start of an additional exposure | 351 (8.2%) | 256 (7.6%) | 584 (8.6%) |
| End of index exposure | 3,344 (78.3%) | 2,674 (79.4%) | 5,277 (78.0%) |
| Maximum follow-up time | 118 (2.8%) | 94 (2.8%) | 205 (3.0%) |
| Specified date reached | 182 (4.3%) | 52 (1.5%) | 270 (4.0%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 169 (4.0%) | 248 (7.4%) | 222 (3.3%) |

• Report overall risk of the primary outcome.

| | Optum CDM | IBM® MarketScan® | CMS - Diabetes | Pooled |
|---|---|---|---|---|
| Risk per 1,000 patients | 25.28 | 12.77 | 31.17 | 25.12 |

#### 8. Initial Power Assessment

#### Aetion report name:

- For Degarelix vs Leuprolide
  - Optum CDM- https://bwh-dope.aetion.com/projects/details/1636/rwrs/67086
  - IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1323/rwrs/67084
  - CMS Diabetes https://bwh-dope.aetion.com/projects/details/1637/rwrs/67082

# Date conducted:

In order to complete the initial power analysis, a dummy outcome indicating a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. A 1:1 PS-matched comparative analysis was performed, including age as the only covariate. Power calculations are based on the formulas

from Chow et al. (2008).

• Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.

Pooled

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 3,934 |
| Reference | 1,967 |
| Exposed | 1,967 |
| Risk per 1,000 patients | 25.12 |
| Desired HR from RCT | 0.49 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 98.82208 |
| Power | 0.943598201 |

Optum CDM

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 1,192 |
| Reference | 596 |
| Exposed | 596 |
| Risk per 1,000 patients | 25.28 |
| Desired HR from RCT | 0.49 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 30.13376 |
| Power | 0.499237002 |

# • IBM® MarketScan®

| Superiority Analysis | |
|----------------------------|------------|
| Number of patients matched | 862 |
| Reference | 431 |
| Exposed | 431 |
| Risk per 1,000 patients | 12.77 |
| Desired HR from RCT | 0.49 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 11.00774 |
| Power | 0.21953525 |

• CMS - Diabetes

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 1,880 |
| Reference | 940 |
| Exposed | 940 |
| Risk per 1,000 patients | 31.17 |
| Desired HR from RCT | 0.49 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 58.5996 |
| Power | 0.779468883 |

Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 3/17/2021 |
|-------------------------|--------------|----------------|-----------|
| Reviewed by FDA: | Ken | Date reviewed: | 4/3/2021 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

# 9. Balance Assessment

# Aetion report name:

# For Degarelix vs. leuprolide

Optum CDM- <a href="https://bwh-dope.aetion.com/projects/details/1636/rwrs/68435">https://bwh-dope.aetion.com/projects/details/1636/rwrs/68435</a>
IBM® MarketScan®- <a href="https://bwh-dope.aetion.com/projects/details/1323/rwrs/68424">https://bwh-dope.aetion.com/projects/details/1323/rwrs/68424</a>

CMS Diabetes - https://bwh-dope.aetion.com/projects/details/1637/rwrs/68434

<u>Date conducted:</u> 04/14/2021

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix\_Table1\_PRONOUNCE\_v1 (worksheet named 'PS matching').

• Report covariate balance after matching.

Note- Please refer to Appendix Table 1 PRONOUNCE v1 (worksheet named 'Table 1').

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Start of an additional exposure | 1147 (30.39%) | 1 (0.05%) | 1146 (60.73%) |
| End of index exposure | 2084 (55.22%) | 1645 (87.18%) | 439 (23.26%) |
| Specified date reached | 157 (4.16%) | 78 (4.13%) | 79 (4.19%) |
| Maximum follow-up reached (365 days) | 142 (3.76) | 42 (2.23%) | 100 (5.30%) |
| End of patient enrollment | 244 (6.46%) | 121 (6.41%) | 123 (6.52%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | | |
|---|---|---|---|
| Patient Group | Optum CDM | IBM® MarketScan® | CMS - Diabetes |
| Overall Patient Population | 89 [64, 116] | 89 [55, 118] | 89 [61, 109] |
| Referent | 89 [89, 89] | 89 [89, 89] | 89 [89, 89] |
| Exposure | 82 [33, 140] | 67 [31, 126] | 68 [33, 125] |

#### **10. Final Power Assessment**

Date conducted: 4/15/2021

Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

#### Pooled

| Superiority Analysis | |
|----------------------------|------------|
| Number of patients matched | 3,774 |
| Reference | 1,887 |
| Exposed | 1,887 |
| Risk per 1,000 patients | 25.12 |
| Desired HR from RCT | 0.49 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 94.80288 |
| Power | 0.93484302 |

## Optum CDM

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 1,092 |
| Reference | 546 |
| Exposed | 546 |
| Risk per 1,000 patients | 25.28 |
| Desired HR from RCT | 0.49 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 27.60576 |
| Power | 0.465815489 |

# • IBM® MarketScan®

| Superiority Analysis | |
|----------------------------|------------|
| Number of patients matched | 830 |
| Reference | 415 |
| Exposed | 415 |
| Risk per 1,000 patients | 12.77 |
| Desired HR from RCT | 0.49 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 10.5991 |
| Power | 0.21311438 |

• CMS - Diabetes

| CIVIS - Diabetes | |
|----------------------------|-------------|
| Superiority Analysis | |
| Number of patients matched | 1,852 |
| Reference | 926 |
| Exposed | 926 |
| Risk per 1,000 patients | 31.17 |
| Desired HR from RCT | 0.49 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 57.72684 |
| Power | 0.773370349 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Date reviewed: |
|-------------------------|----------------|
| Reviewed by FDA: | Date reviewed: |
| Reasons for stopping | |
| analysis (if required): | |

# 11. Study Confidence and Concerns

Deadline for voting on study confidence and listing concerns:

Date votes and concerns are summarized:

• If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.

- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the success of the RWD study in the <a href="Google Form">Google Form</a>. This form also provides space for reviewers to list any concerns that they feel may contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the individual respondent.
- After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

#### 12. Register study protocol on clinicalTrials.gov

Date conducted:

• Register the study on clinicalTrials.gov and upload this document.

#### 13. Comparative Analyses

Aetion report name:

Date conducted:

- 13.1 For primary analysis:
- 13.2 <u>For sensitivity analyses:</u>

# 14. Requested Results

#### 14.1 Table 1: Baseline characteristics before and after adjustment

| Variable | Before adjustment | | | After adjustment | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |

# 14.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

# 14.3 <u>Table 3: Censoring events</u>

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

# 14.4 <u>Table 4: Results from primary analyses;</u>

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

# 14.5 <u>Table 5: Results from secondary analyses;</u>

# 15. References

Chow S, Shao J, Wang H. 2008. *Sample Size Calculations in Clinical Research*. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

# Appendix A

# **Information from Trial**

<u>Trial Name:</u> PRONOUNCE https://www.clinicaltrials.gov/ct2/show/NCT02663908

NCT: NCT02663908

Therapeutic Area: Oncology

**RCT Category:** Equivalence/Superiority

**Brand Name:** Firmagon

**Generic Name:** Degarelix

**Sponsor:** Ferring Pharmaceuticals

Year: 2016 - Present

**Measurable Endpoint:** MACE

Exposure: Degarelix

**Comparator:** Leuprolide

**Populuation:** Men of any age with with advance prostate cancer and predefined CV disease

No. of Patients: TBD

**Power:** TBD

# Appendix A

| | PRONOUNCE trial definitions | Implementation in routine care | | Out on a disco |
|---|---|---|---|---|
| <u>-</u> | PRONOUNCE trial definitions | *************************************** | References/Rationale Please see the following Google Drive for further details or any missing information: | Color coding |
| | | TRIAL DETAILS | Please see the following Google Drive for further details or any missing information:<br>https://drive.google.com/open?id=1WD618wnywYjEAXrll.TcuK-VCcnb6b-gV | Criteria |
| 1 | | | ICD-10 codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be available in the above Google Drive Fulder (link above) ICD-8 to ICD-10 code conversions. | |
| 1 | | | Full ICO-10 code lists will be available in the above Google Prive Folder films abovels ICO-2 to ICO-10 code conversions;<br>axes completed using a SAS macro that implements forward! backward mapping based on the CNS ICO-9 to ICO-10<br>mapping; this prive window or or glossal icd9 -cd-10 cm -and price-rosswalls general -equivalence mapping html | |
| | | EXPOSURE vs. COMPARISON | париц, поредникалин от рован получен зочения усектомние унив в черочивное парушулин | Can be replicated in claims |
| vs. | 1 month, Degarelix 80mg SC q mt x 11 months thereafter | <u>Degarelix Arm</u> : Generic name: Degarelix Acetate; HCPCS/CPT: J915S (inpatient and outpatient) vs. | | Using dummy definitions for measuring in claims |
| Leuprolide IM 22.5mg q 3 mc | months x 12 months | Leuprolide Arm: Generic name: Leuprolide Acetate; HCPCS/CPT: J1950, C9430, J9219, J9218, J9217 (inpatient and outpatient) | | Can't he measured in claims |
| | | Measured from first day following expoure initiation | | |
| | | Death: Inpatient death indicated by discharge date | | |
| | | Seafort Mic 70 - Slagonic - 416 to GETF - 410.2 20 - 50 - 50 - 50 - 50 - 50 - 50 - 50 - | | |
| MACE (All-cause death, nonfatal | tal myocardial infarction, nonfatal stroke) | Norfatal Stroke: Stroke (ischemic/hemorrhagic): ICD-9 diagnosis: "430", "431", "433.01", "433.11", "433.31", "433.31", "433.91", "434.01", "434.01", "434.01", "434.01", "434.11", "434.91", "436.00", "431", "435.00", "431", "433.01", "43 | Source: CANVAS trial (https://bwh-dope.aetion.com/measures/details/92945/661/0/basics) | Can't be measured in claims but not important for the analysis |
| | | \$5.09 \$63.00 \$63.01 \$63.02 \$63.09 \$63.00 \$63.01 \$63.11 \$63.12 \$63.19 \$63.19 \$63.10 \$63.11 \$63.12 \$63.19 \$63.10 \$63.11 \$63.12 \$63.19 \$63.19 \$63.10 \$63.11 \$63.12 \$63.19 \$63.10 \$63.11 \$63.12 \$63.19 \$63.10 \$63 | | |
| | | 63.511 (63.512 (63.512) (63.521 (63.523 (63.523 (63.531 (63.532 (63.539 (63.541 (63.542 (63.546 (63.54 | | |
| | | INCLUSION CRITERIA | | |
| | | Measured from (start of all available data, 0). Must have both, diagnosis code and male gender for inclusion. | Male patients with 1 dx code + an exposure provides enough information to confirm diagnosis, as the<br>exposures have very few or no indications outside of advanced PC | |
| 1 Histologically confirmed ade | denocarcinoma of the prostate | Malignant Neoplasm of the Prostate:<br>ICD 9 diagnosis: 185:xxx | Necessitating code for biopsy may exclude subjects with prevalent prostate cancer if they were initially | |
| | | ICD-10 diagnosis; C61.x (inpatient and outpatient) | diagnosed prior to database enrollment with early stage disease | |
| | | See: Male | Lupron is indicated in females for endometriosis. Restricting to males helps ensure indication of interest. | |
| Tumor, node, metastasis staj<br>study start | taging available before treatment start (bone scan and/or CT scan and/or MRI) <12 weeks before | | | |
| | initiate continued ADT therapy with intended duration of 12 months or longer | | | |
| -Patients with metastatic | initiate continued ADT therapy with intended duration of 12 months or longer<br>is prostate cancer at time of diagnosis<br>cancer who develop metastases after local therapy<br>cancer with very high-risk, high-risk, or intermediate risk disease with feature of unfavorable<br>edw who definiter readiation therapy in combination with at least 12 months of | | | |
| Patients with prostate ca | cancer with very high-risk, high-risk, or intermediate risk disease with feature of unfavorable | | | |
| prognosis who will be treate-<br>neoadjuvant/adjuvant ADT | ted with definitive radiation therapy in combination with at least 12 months of | | | |
| | | Measured from [start of all available data , -30] in an inpatient or outpatient care setting in any diagnosis position | | |
| Pre-existing ASCAID (co-fr- | med diagnosis, documented) according to at least 1 of the following criteria. | Acute or old MI: | | |
| -Previous myocardial infa | med diagnosis, documented) according to at least 1 of the following criteria<br>farction >= 30 days before randomization | SCD-9 disagnosis: 410.xx , 412.xx<br>SCD-10 disagnosis: 121.01, 121.02, 121.09, 121.11, 121.19, 121.21, 121.29, 121.3, 121.4, 122.0, 122.1, 122.2, 122.8, 122.9, 125.2 | | |
| Previous revascularizatio Coronary artery: stent pli | ion procedure >=30 days before randomization<br>placement/balloon angioplasty or coronary artery bypass graft surgery | Company of the Company Company of the Company of th | Sources: DUPLICATE Standard Measures ("MI (Inc3 HF Algorithm)", "Old MI with ICD 10 Copy") | |
| <ul> <li>Carotid artery: stent place</li> <li>Iliac, femoral, popliteal</li> </ul> | olacement/balloon angioplasty or coronary artery bypass graft surgery<br>acement/balloon angioplasty or endarterectomy surgery<br>arteries: stent placement/balloon angioplasty or vascular bypass surgery | (CD-9 procedure: "00.66", "36.03", "36.06", "36.07", "36.09", "36.13", "36.32", "36.33", "36.34", "36.10", "36.11", "36.12", "36.13", "36.14", "36.15", "36.16", "36.16", "36.16", "36.16", "36.16", "36.17", "36.18", "36. | | |
| | | ICD-10 procedure: see Appendix HEPCS/(PT: "35302", "35356", "35363", "35372", "35372", "35381", "35483", "35483", "35521", "35533", "35539", "35540", "35540", "35540", "35540", "35549", "35551", "35555", "35556", "35556", "35565", "35665", "35665 | DUPLICATE Standard Measures ("Old MI with ICD 10 Copy", "Information on Outcome- Coronary revascularization (PTCA, stenting, CABG) v5 -WITH ICD-10 CODES") | |
| | | "35646", "35651", "35651", "35656", "35666", "35665", "35666", "35666", "34201", "34203", "34421", "34451", "35303", "35571", "35623", "35671" | revascularization (PTCA, stenting, CABG) v5 -WITH ICD-10 CODES") | |
| -Coronany arteny | >=50% at any time point before randomization by angiography or CT angiography | | | |
| Carotid artery Iliac, femoral, or poplite | eal arteries | | | |
| -Carotid ultrasound result | eal arteries Its that documented a vascular stenosis >=50% at any time point before randomization Index <0.9 at any time point before randomization | | | |
| | and the same part of the same same same same same same same sam | EXCLUSION CRITERIA | | |
| | | Measured [-365, 0] in an inpatient or oupatient care setting in any diagnosis position | | |
| Patients must be treatment- | t-naive (ADT) | GriPRI Agonists: generic name: goverelin; triptorelin; histrelin: HEPCS/CPT: goverelin: 19202 59560; triptorelin: 13315 13315 histrelin: 11675 19225 19226 0,2020 50133 (inpatient and outpattent) | Source:https://jamanetwork.com/journals/jamaoncology/article-abstract/2476248 | |
| 1 months before randomizatio | ion | Measured (-365, -14) | Patients may fill prescription and initiate androgen blockade ~1-2 weeks prior to start of LHRH agonist for flare | |
| <ul> <li>Any additional hormonal<br/>initial flare protection is allo</li> </ul> | toware (unit) folious ADT for necadjuvant or adjuvant therapy, then the last dose of therapy must be at least 12 ion at herapy upfront (i.e., abiraterone) is prohibited in the study, however, anti-androgen use for owed for a maximum period of up to 28 days after randomization | | protection | |
| | | Harmonal Therapy: generic name: abiraterone, ketoconazole, flutamide, bicalutamide, nilutamide, enzalutamide, apalutamide, finasteride, dutasteride<br>HEPCS/COT: flutamide: 50175 finasteride: 50138 | | |
| | | Measured from (start of all available data , 0) in an inpatient and outpatient care setting in any diagnosis position: | | |
| | | Orchiectomy: HCPCS/CPT: 54520, 54522, 54530, 54535, 54690 (54521 not found in databases) | | |
| | | CD-9 procedure: 62.3x, 62.4x (Inpatient and outpatient) CD-10 procedure: "0VT90ZZ", "0VT94ZZ", "0VT84ZZ", "0VTC0ZZ", "0VTC0ZZ" | Source:https://jamanetwork.com/journals/jamaoncology/article-abstract/2476248 | |
| Previous or current hormonal | ial management of prostate cancer | Measured [-365, 0]: | patients may initiate androgen blockade for flare within 14 days of initial treatment, which is permissible per | |
| Surgical castration Any hormonal manipulati | ation | GRRH Agoelsts: generic name: goserelin, triptorelin, histrelin | PRONOUNCE selection criteria | |
| | ant/adjuvant hormonal therapy, unless treatment terminated >12 months before study start | ICPCS/CPT: gonerellin: 19202 59560; triptorellin: 13315 13316 histrellin: 11675 19225 19226 Q2020 50133 (inpatient and outpatient) | Abarelix was not included, as it was only on the market for a short period of time prior to the span of our data resources. Cetrorelix and ganirelix are also excluded from this analysis since they're not indicated for prostate | |
| | | Measured (-365, -14): | cancer. | |
| | | Hormonal Therapy: generic name: abiraterone, ketoconazole, flutamide, bicalutamide, nilutamide, enzalutamide, apalutamide, finasteride, dutasteride | | |
| | | HEPCS/CPT: flutamide: S0175 finasteride: S0138 | | |
| | | Measured [-30, 0] in an inpatient care setting in a primary diagnosis position | | |
| | | Uncontrolled Diabetes | L | |
| 3 Uncontrolled type 1 or type | | ICD-9: 790.29 | Source: Lodes from Duplicate standard measure library (https://bwn- | |
| ,, == 1,,== | 2 diabetes mellitus (defined as HbA1c >10%) at time of randomization | <u>KD-10.</u> R73.09, R73.9 | Source: Codes from Duplicate standard measure library (https://bwh-<br>dope.aetion.com/measures/details/306630/0/0/templates/simpleEventSet?tab=3) | |
| | 2 diabetes mellitus (defined as HbAIc >10%) at time of randomization | <u>500-2</u> 70-23<br><u>500-10</u> (77.00, 873-9 | An inpatient, primary diagnosis of hyperglycemia is thought to be a good proxy for uncontrolled diabetes based | |
| | 2 diabetes mellitus (defined as HbA1c >10%) at time of randomization | <u>509-2</u> 70.29<br><u>509-0</u> 773.00, 873.9 | | |
| | 2 diabetes mellitus (defined as HbALc >10%) at time of randomization | <u>550 10</u> 872.09, 872.9 | An inpatient, primary diagnosis of hyperglycemia is thought to be a good proxy for uncontrolled diabetes based | |
| | 2 diabetes mellitus (defined as HRA1: >10%) at time of randomization | 202.10, F72.00, R72.9 Measured 30, 0] (CD-10 measured in other an inpatient or outpatient care setting in any diagnosis position. ICD-9 measured in an inpatient care setting or ED setting in a primary diagnosis position: | An inpatient, primary diagnosis of hyperglycemia is thought to be a good proxy for uncontrolled diabetes based | |
| | | 202.10, F72.00, R72.9 Measured 30, 0] (CD-10 measured in other an inpatient or outpatient care setting in any diagnosis position. ICD-9 measured in an inpatient care setting or ED setting in a primary diagnosis position: | An inpatient, primary diagnosis of hyperglycemia is thought to be a good proxy for uncontrolled diabetes based | |
| 4 Uncontrolled hypertension (S | 2 diabetes mellitus (defined as HBALs >10%) at time of randomization (SBP >180 mm Hg or OBP >110 mm Hg) at time of randomization | <u>550 10</u> 872.09, 872.9 | An inpatient, primary diagnosis of hyperglycemia is thought to be a good proxy for uncontrolled diabetes based | |
| 4 Uncontrolled hypertension (S | | 202.10, F72.00, R72.9 Measured 30, 0] (CD-10 measured in other an inpatient or outpatient care setting in any diagnosis position. ICD-9 measured in an inpatient care setting or ED setting in a primary diagnosis position: | An inpatient, primary diagnosis of hyperglycennia is thought to be a good proxy for uncontrolled diabetes based<br>on the investigation's selectative knowledge. | |
| 4 Uncontrolled hypertension (\$ | | 202.10, F72.00, R72.9 Measured 30, 0] (CD-10 measured in other an inpatient or outpatient care setting in any diagnosis position. ICD-9 measured in an inpatient care setting or ED setting in a primary diagnosis position: | An inpatient, primary diagnosis of hyperglycemia is thought to be a good proxy for uncentrolled diabetes based on the investigation's additional knowledge. Source: CUPLICATE Team (EMPEROR-Presenced trial) | |
| 4 Uncontrolled hypertension (S | | ISO 10: 173.09, 873.9 Measured [ 35, 6] CD-1D measured in other an inpatient or outpatient care setting in any diagnosis position. CD-5 measured in an inpatient care setting or CD setting in a primary diagnosis position. Soliganest hypertension/Hypertension/CD-10. Soliganest hypertension/Hypertension/Hypertension/CD-10. Soliganest hypertension/Hypertension/CD-10. Soliganest hypertension/Hypertension/Hypertension/CD-10. Soliganest hypertension/Hypertension/CD-10. Soliganest hypertension/Hypertension/Hypertension/CD-10. Soliganest hypertension/Hy | An inpatient, primary diagnosis of hyperglycemia is thought to be a good proxy for uncentrolled diabetes based on the investigation's additional knowledge. Source: CUPLICATE Team (EMPEROR-Presenced trial) | |
| 4 Uncontrolled hypertension (5 | | 20.10. F73.05, 6729 Measure[ 30, 0] CD-1D measured in other an inpatient or outpatient care setting in any diagnosis position. KD-9 measured in an inpatient care setting or ED setting in a primary diagnosis position: Measure[ 150, 0] KD-1D measured in other an inpatient or outpatient care setting in any diagnosis position. KD-9 measured in an inpatient care setting or ED setting in a primary diagnosis position: 86.0 8 4 4 4 4 5 5 5 5 6 4 4 4 5 5 5 5 6 6 6 6 | An inpatient, primary diagnosis of hyperglycemia is thought to be a good proxy for uncentrolled diabetes based on the investigation's additional knowledge. Source: CUPLICATE Team (EMPEROR-Presenced trial) | |
| 4 Uncontrolled hypertension (s | | Each 10, 173.00, 172.9 Measured [34, 6] CD-10 measured in either an inpatient or outpatient care setting in any diagnosis position. ICD-9 measured in an inpatient care setting or ID setting in a primary diagnosis position. Measured [34, 6] CD-10 measured in either an inpatient or outpatient care setting in any diagnosis position. Measured [34, 6] CD-10 measured in an inpatient care setting in a primary diagnosis position. Measured [34, 6] CD-10 measured in either an inpatient care setting in any diagnosis position. Local diagnosis [35, 6] CD-10 measured in either an inpatient care setting in any diagnosis position. Local diagnosis [35, 6] CD-10 measured in either an inpatient or outpatient care setting in any diagnosis position. Local diagnosis [35, 6] CD-10 measured in either an inpatient or outpatient or outpatient care setting in any diagnosis position. Local diagnosis [35, 6] CD-10 measured in either an inpatient or outpatient or outpatient care setting in any diagnosis position. | An inpatient, primary diagnosis of hyperglycemia is thought to be a good proxy for uncentrolled diabetes based on the investigation's additional knowledge. Source: CUPLICATE Team (EMPEROR-Presenced trial) | |
| 4 Uncontrolled hypertension (5 | | CO.10. 177.00, 872.9 Measured (34, 0) (CO-10 measured in either an inpatient or outpatient care setting in any diagnosis position. XCD-9 measured in an inpatient care setting or ID setting in a primary diagnosis position. Measured (34, 0) (CO-10 measured in either an inpatient or outpatient or outpatient care setting in any diagnosis position. Measured (34, 0) (CO-10 measured in either an inpatient care setting in a primary diagnosis position. Measured (34, 0) (CO-10 measured in either an inpatient care setting in any diagnosis position. Measured (34, 0) (CO-10 measured in either an inpatient care setting in any diagnosis position. Measured (34, 0) (CO-10 measured in either an inpatient care setting in any diagnosis position. Measured (34, 0) (CO-10 measured in either an inpatient care setting in any diagnosis position. Measured (34, 0) (CO-10 measured in either an inpatient care setting in any diagnosis position. Measured (34, 0) (CO-10 measured in either an inpatient care setting in a primary diagnosis position. Measured (34, 0) (CO-10 measured in either an inpatient care setting in a primary diagnosis position. Measured (34, 0) (CO-10 measured in either an inpatient care setting in any diagnosis position. Measured (34, 0) (CO-10 measured in either an inpatient care setting in an inpatient care setting in a primary diagnosis position. Measured (34, 0) (CO-10 measured in either an inpatient care setting in a primary diagnosis | An inpatient, primary diagnosis of hyperglycemia is thought to be a good proxy for uncentrolled diabetes based on the investigation's additional knowledge. Source: CUPLICATE Team (EMPEROR-Presenced trial) | |
| Uncontrolled hypertension () | | Example (19, 6) (CD-10 measured in either an inpatient or outpatient cure setting in any diagnosis position XCD-9 measured in an inpatient cure setting or ID setting in a primary diagnosis position. Molignant hypotrension/Hypotrension/ | An inpatient, primary diagnosis of hyperglycemia is thought to be a good proxy for uncentrolled diabetes based on the investigation's additional knowledge. Source: CUPLICATE Team (EMPEROR-Presenced trial) | |
| | (SBP > 180 mm Hg or OBP > 110 mm Hg) at time of randomization | 66-saured [36, 6] CD-10 measured in either an inpatient or outpatient care setting in any diagnosis position. KD-9 measured in an inpatient care setting or ID setting in a primary diagnosis position. Malignatis Appartantion/Repertantions cable. 60-5 Bearmonia, 916, 92.11, 401.2, 401.0, 401.0, 404.0, 405.0, 401.9, 417.2, 796.2 CD-10 diagnosis; 164.8 60-6 Saured [1st of all available data, 0] in an inpatient or outpatient care setting in any diagnosis position Long CE Syndrome: CD-9 saured [1st of all available data, 0] in an inpatient or outpatient care setting in any diagnosis position Long CE Syndrome: CD-9 saured [1st, 0] in a limpatient code or outpatient codes in any diagnosis position Measured [36, 6] in a limpatient code or outpatient codes in any diagnosis position Long CE Syndrome: CD-9 saured [1st, 0] in a limpatient code or outpatient codes in any diagnosis position Long CE Syndrome; CD-9 saured [1st, 0] in a limpatient code or outpatient codes in any diagnosis position Long CE Syndrome; CD-9 saured [1st, 0] in a limpatient code or outpatient codes in any diagnosis position Long CE Syndrome; CD-9 saured [1st, 0] in a limpatient code or outpatient codes in any diagnosis position Long CE Syndrome; CD-9 saured [1st, 0] in a limpatient code or outpatient codes in any diagnosis position Long CE Syndrome; CD-9 saured [1st, 0] in a limpatient code or outpatient codes in any diagnosis position Long CE Syndrome; CD-9 saured [1st, 0] in a limpatient code or outpatient codes in any diagnosis position Long CE Syndrome; CD-9 saured [1st, 0] in a limpatient code or outpatient codes in any diagnosis position Long CE Syndrome; CD-9 saured [1st, 0] in a limpatient code or outpatient codes in any diagnosis position Long CE Syndrome; CD-9 saured [1st, 0] in a limpatient code or outpatient codes in any diagnosis position Long CE Syndrome; CD-9 saured [1st, 0] in a limpatient code or outpatient codes in any diagnosis position Long CE Syndrome; CD-9 saured [1st, 0] in a limpatient code or o | An inpatient, primary diagnosis of hyperglycennia is thought to be a good proxy for uncontrolled diabetes based on the investigation's selectation knowledge. Source: CUPILCATE Team (IMPEROR Preserved trial) Malignant HTM clinically defined as SBP-180mmitg Source: CUPILCATE Standard Measure ("Heart Failure (CHF) Ever Lookback"), CMED Measure Library | |
| A Niction of connected loss of | (SBF > 180 mm lig or OBF > 110 mm lig) at time of randomization | Measured [34, 0] (CD-10 measured in either an inpatient or outpatient care setting in any diagnosis position. XCD-9 measured in an inpatient care setting or ID setting in a primary diagnosis position. Measured [34, 0] (CD-10 measured in either an inpatient or outpatient care setting in any diagnosis position. Measured [34, 0] (CD-10 measured in either an inpatient or outpatient or outpatient care setting in any diagnosis position. Measured [34, 0] (CD-10 measured in either an inpatient or outpatient care setting in any diagnosis position. Measured [34, 0] (CD-10 measured in either an inpatient care setting in any diagnosis position. Measured [34, 0] in an inpatient code or 2 outpatient code in any diagnosis position. Measured [34, 0] in an inpatient code or 2 outpatient code in any diagnosis position. CD-10 diagnosis (24, 28, 38, 34, 4021, 4031, 4031, 4041, 4041, 4043); CD-10 diagnosis (24, 28, 38, 34, 4021, 4031, 4031, 4041, 4043); CD-10 diagnosis (24, 28, 38, 34, 4021, 4031, 4031, 4041, 4043); CD-10 diagnosis (24, 28, 38, 34, 4021, 4031, 4031, 4041, 4043); CD-10 diagnosis (24, 28, 38, 34, 4021, 4031, 4031, 4041, 4043); CD-10 diagnosis (24, 28, 34, 4041, 4041, 4041, 4043); CD-10 diagnosis (24, 38, 34, 4041, 4041, 4043); CD-10 diagnosis (24, 38, 34, 4041, 4041, 4043); CD-10 diagnosis (24, 38, 34, 4041, 4041, 4041, 4043); CD-10 diagnosis (24, 38, 34, 4041, 4041, 4041, 4041, 4043); CD-10 diagnosis (24, 38, 34, 4041, 4041, 4041, 4043); CD-10 diagnosis (24, 38, 34, 4041, 4041, 4041, 4041, 4041, 4041, 4041); CD-10 diagnosis (24, 34, 34, 4041, 4 | an installed, primary diagnosis of hyperplycensis is thought to be a good proxy for uncontrolled diabetes based on the investigators' substantive knowledge. Source: OUPLICATE Team (EMPEROR-Preserved trial) Malignant HTM clinically defined as \$899-130mmitg Source: OUPLICATE Standard Measure ("Heart Failure (OH) Ever Lookback"); ORIO Measure Library ("REPAT, Redact, 13), OT Polloging drugs"). Aerion Santh, Aerion Search | |
| A history of connectival loss of | (SBP > 180 mm Hg or OBP > 110 mm Hg) at time of randomization | Measured [30, 0] (CD-10 measured in other an inpatient or outpatient care setting in any diagnosis position. ICD-9 measured in an inpatient care setting or ID setting in a primary diagnosis position. Maligneth Physitemetric Physitemetric Physitemetric Care Setting in any diagnosis position. ICD-9 measured in an inpatient care setting or ID setting in a primary diagnosis position. Maligneth Physitemetric Physitemetric Care Setting in any diagnosis position. Measured [316, 0] (CD-10 measured diata, 0] in an inpatient or outpatient care setting in any diagnosis position. Measured [316, 0] (CD-10 measured diata, 0] in an inpatient or outpatient care setting in any diagnosis position. Measured [316, 0] (CD-10 measured diata, 0] in an inpatient code or a outpatient care setting in any diagnosis position. Measured [316, 0] (CD-10 measured diata, 0] in an inpatient code or 2 outpatient codes in any diagnosis position. Measured [316, 0] (CD-10 measured diata, 0] in an inpatient code or 2 outpatient codes in any diagnosis position. Measured [310, 0] (CD-10 measured diata, 0] in an inpatient code or 2 outpatient codes in any diagnosis position. Measured [310, 0] (CD-10 measured diata, 0] in an inpatient code or 2 outpatient codes in any diagnosis position. Measured [310, 0] (CD-10 measured diata, 0] in an inpatient code or 2 outpatient codes in any diagnosis position. Measured [310, 0] (CD-10 measured diata, 0] in an inpatient code or 2 outpatient codes in any diagnosis position. Measured [310, 0] (CD-10 measured diata, 0] in an inpatient code or 2 outpatient codes in any diagnosis position. Measured [310, 0] (CD-10 measured diata, 0] in an inpatient code or 2 outpatient codes in any diagnosis position. | an installed, primary diagnosis of hyperplycensis is thought to be a good proxy for uncontrolled diabetes based on the investigators' substantive knowledge. Source: OUPLICATE Team (EMPEROR-Preserved trial) Malignant HTM clinically defined as \$899-130mmitg Source: OUPLICATE Standard Measure ("Heart Failure (OH) Ever Lookback"); ORIO Measure Library ("REPAT, Redact, 13), OT Polloging drugs"). Aerion Santh, Aerion Search | |
| A history of connectival loss of | (SBF > 180 mm lig or OBF > 110 mm lig) at time of randomization | Measured (34, 6) (CD-10 measured in either an injustient or outpatient care setting in any diagnosis position KD-9 measured in an injustient care setting or ID setting in a primary diagnosis position KD-9 measured in an injustient care setting or ID setting in a primary diagnosis position KD-9 measured in an injustient care setting or ID setting in a primary diagnosis position KD-9 measured in an injustient care setting in any diagnosis position in an injustient care setting in any diagnosis position in any diagnosis position in any diagnosis position in an injustient code or 2 outpatient codes in any diagnosis position in | An inpatient, primary diagnosis of hyperglycennia is thought to be a good proxy for uncontrolled diabetes based on the investigation's selectation knowledge. Source: CUPILCATE Team (IMPEROR Preserved trial) Malignant HTM clinically defined as SBP-180mmitg Source: CUPILCATE Standard Measure ("Heart Failure (CHF) Ever Lookback"), CMED Measure Library | |
| A history of connectival loss of | (SBF > 180 mm lig or OBF > 110 mm lig) at time of randomization | Measured [30, 8] CD-10 measured in other an inputient or outpatient care setting in any diagnosis position. XCD-9 measured in an inputient care setting or ID setting in a primary diagnosis position. Measured [30, 8] CD-10 measured in inputient or outpatient care setting in any diagnosis position. XCD-9 measured in an inputient care setting or ID setting in a primary diagnosis position. Measured [30, 8] CD-10 measured in an inputient or outpatient care setting in any diagnosis position. Measured [31, 8] CD-10 measured data, g) in an inputient or outpatient care setting in any diagnosis position. Measured [31, 8] (a) in a Linguistic code or 2 outpatient codes in any diagnosis position. Measured [31, 8] (a) in an Linguistic code or 2 outpatient code outpatie | an installed, primary diagnosis of hyperplycensis is thought to be a good proxy for uncontrolled diabetes based on the investigators' substantive knowledge. Source: OUPLICATE Team (EMPEROR-Preserved trial) Malignant HTM clinically defined as \$899-130mmitg Source: OUPLICATE Standard Measure ("Heart Failure (OH) Ever Lookback"); ORIO Measure Library ("REPAT, Redact, 13), OT Polloging drugs"). Aerion Santh, Aerion Search | |
| A history of commonly loop of | (SBF > 180 mm lig or OBF > 110 mm lig) at time of randomization | Measured [30, 0] ICD-1D measured in other an inpatient or outpatient care setting in any diagnosis position. ICD-9 measured in an inpatient care setting or ID setting in a primary diagnosis position. Moligonath inpatient (AD-9 measured in an inpatient care setting in a primary diagnosis position. ICD-9 measured in an inpatient care setting in a primary diagnosis position. Moligonath inpatient of all availables data, 0] in an inpatient or outpatient care setting in any diagnosis position. Moligonath inpatient of all availables data, 0] in an inpatient or outpatient care setting in any diagnosis position. Moligonath inpatient of all availables data, 0] in an inpatient or outpatient care setting in any diagnosis position. Moligonath inpatient of all availables data, 0] in an inpatient code or 2 outpatient codes in any diagnosis position. Moligonath inpatient code or 2 outpatient codes in any diagnosis position. Moligonath inpatient code or 2 outpatient codes in any diagnosis position. Moligonath inpatient code or 2 outpatient codes in any diagnosis position. Moligonath inpatient codes or 2 outpatient codes in any diagnosis position. Moligonath inpatient codes or 2 outpatient codes in any diagnosis position. Moligonath inpatient codes or 2 outpatient codes in any diagnosis position. Moligonath in an inpatient code of 2 outpatient codes in any diagnosis position. Moligonath in an inpatient code of 2 outpatient codes in any diagnosis position. Moligonath in an inpatient code of 2 outpatient codes in any diagnosis positio | an installed, primary diagnosis of hyperplycensis is thought to be a good proxy for uncontrolled diabetes based on the investigators' substantive knowledge. Source: OUPLICATE Team (EMPEROR-Preserved trial) Malignant HTM clinically defined as \$899-130mmitg Source: OUPLICATE Standard Measure ("Heart Failure (OH) Ever Lookback"); ORIO Measure Library ("REPAT, Redact, 13), OT Polloging drugs"). Aerion Santh, Aerion Search | |
| A history of commonly loop of | (SBF > 180 mm lig or OBF > 110 mm lig) at time of randomization | Measured [54, 6] (CD-10 measured in either an inpatient or outpatient care setting in any diagnosis positionKD-9 measured in an inpatient care setting or ED setting in a primary diagnosis position. Molignant Proportion Mayorization (Hypertacobia) cubic 50 6 aleganesis (45) a. 80.21.1. 401.0. 402.0., 403.0., 403. | an installed, primary diagnosis of hyperplycensis is thought to be a good proxy for uncontrolled diabetes based on the investigators' substantive knowledge. Source: OUPLICATE Team (EMPEROR-Preserved trial) Malignant HTM clinically defined as \$899-130mmitg Source: OUPLICATE Standard Measure ("Heart Failure (OH) Ever Lookback"); ORIO Measure Library ("REPAT, Redact, 13), OT Polloging drugs"). Aerion Santh, Aerion Search | |
| A history of connentral loop ( | (SBF > 180 mm lig or OBF > 110 mm lig) at time of randomization | Measure [ 30, 8] CD-10 measured in other an inpatient or outpatient care setting in any diagnosis position. XD-9 measured in an inpatient care setting or ID setting in a primary diagnosis position. Measure [ 30, 8] CD-10 measured in an inpatient or outpatient care setting in any diagnosis position. XD-9 measured in an inpatient care setting or ID setting in a primary diagnosis position. Measured [ 15, 10, 10 | an installed, primary diagnosis of hyperplycensis is thought to be a good proxy for uncontrolled diabetes based on the investigators' substantive knowledge. Source: OUPLICATE Team (EMPEROR-Preserved trial) Malignant HTM clinically defined as \$899-130mmitg Source: OUPLICATE Standard Measure ("Heart Failure (OH) Ever Lookback"); ORIO Measure Library ("REPAT, Redact, 13), OT Polloging drugs"). Aerion Santh, Aerion Search | |

# Appendix A

| 6 | Within 30 days before randomination: Application infection -trainel (hemorrally circlemic) -coronary, carotid, or peripheral artery revascularization | DUPLICATE Standard Measure ("Information on Outcome - Stroke WITH ICD-10 CODES [Inpatient, PRIMARY)", "Acute Mil [INVER LODING ACQ[")"] |
|---|---|---|
| 7 | Planned or scheduled cardiac surgery or PCI procedure that is known at the time of randomization | |



# Table 1 Unmatched

| Company Comp | | | | UNMA | TCHED | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Name | | | | | | | Medicare Pool | | | | | | oled |
| Text of Confect Control (1997) 1. | Variable | Leuprolide | | St. Diff | Leuprolide | Degarelix | St. Diff | Leuprolide | Degarelix | St. Diff | Leuprolide | Degarelix | St. Diff |
| 2005.0701 1907.0702 1907.0703 1907 | Number of patients | 3,681 | 597 | | 2,938 | 431 | | 5,829 | 941 | | 12,448 | 1,969 | |
| 2001 1 PM | Year of Cohort Entry Date | | | | | | | | | | | | |
| 2011 - (N) | 2008-2009; n (%) | 262 (7.1%) | - ( / | | | 0 (0.0%) | 0.49 | 353 (6.1%) | - ( / | 0.36 | 927 (7.4%) | - ( / | |
| 2011-101 245-57 241-57 2 | | | | | | | | | | | | | |
| | | | , , | | | | | | | | | | |
| 2.255.e. (h) | | | , , | | | | | | | | | | |
| 2,351 f. n/s) | | | , , | | | | | | | | | | |
| 2016.4 | | | , , | | | | | . , | | | , , | | |
| 2,301 a. NS | | | | | | | | | | | | | |
| | | | | | | | | . , | | | | | |
| 2.2026 n/N 47911360 30107.3% 0.012 | | | | | | | | | 169 (18.0%) | -0.19 | 1,251 (10.0% | 297 (15.1%) | -0.15 |
| | | | | | 114 (3.9%) | 27 (6.3%) | -0.11 | | | | | | |
| Age Company | | | . , | | | | | | | | | | |
| men (pd) | | 265 (7.2%) | 40 (6.7%) | 0.02 | | | | | | | | | |
| media pi(i) 76.00 7.00 7.00 7.00 7.00 8.00 7.00 7.00 8.00 7.00 | | 75 74 /7 42) | 75 02 (7 65) | 0.03 | 74 20 (0.05) | 74.40 (0.42) | 0.01 | 76.05 (6.50) | 76.04 (6.40) | 0.01 | 75 02 (7 40) | 76 40 (7 40) | 0.03 |
| Nether 10 36 (6 9 %) 9 16 (6 %) 0.00 22 16.4 % 9 12 (2 %) 0.00 1.00 | ` ' | . , | , , | | | | | | | | | | |
| 1.4 Post Protecting (19) | | / 0.00 [/1.00, | 70.00 [71.00] | 0.00 | 75.00 JU.61 | , 75.00 [08.00] | , 0.00 | 70.00 [72.00, | 77.00 [72.00, | -0.15 | 75.70 (8.86) | /0.20 (8.81) | -0.06 |
| 2 North Central, (Ps) | | 366 (9 0%) | 99 (16 6%) | -n 2n | 423 (14 49/) | 95 (22 0%) | -n 2n | 1 018/17 50/ | 194 (20 6%) | _n no | 1 807 /14 = 0/ | 388 (10 70/1 | -0.14 |
| | | | | | , , | | | | | | , , | | |
| New | | | | | | | | | | | | | |
| | | 323 (23.170) | 131 (21.370) | 0.00 | 420 (14.570) | 45 (11.470) | 0.03 | 300 (10.370) | 147 (15.070) | 0.04 | 2,555 (10.770 | 327 (10.070) | 0.00 |
| Asian; (%) | | 2.727 (74.1%) | 448 (75.0%) | -0.02 | | | | 4.818 (82.7% | 806 (85.7%) | -0.08 | 7.545 (60.6% | 1.254 (63.7% | -0.06 |
| Black n (N) | | | | | | | | | | | | | _ |
| Hispanic, (16) | | | , , | | | | | | | | | | |
| | | | | -0.01 | | | | | | | | | |
| Cardiovascular event prognosticators | North American Native; n (%) | | | | | | | N/A | N/A | N/A | N/A | N/A | N/A |
| Acute or Old Mr.; (%) 1.428 (8.8.8%) [232 (8.9.9%) | Other; n (%) | | | | | | | 108 (1.9%) | 16 (1.7%) | 0.02 | 108 (1.9%) | 16 (1.7%) | 0.02 |
| Anxiety, n(s) Anxiet | Cardiovascular event prognosticators | | | | | | | | | | | | |
| Attrial Fibrillation; n (%) Coronary, Attrial Fibrillation; n (%) Coronary, Carotid, Illiac, Femoral, and Popitiea Revascularization (Angioplasty/Stent/CABS); n (38, 18, 19, 19, 10) Coronary, Carotid, Illiac, Femoral, and Popitiea Revascularization (Angioplasty/Stent/CABS); n (38, 18, 19, 19, 10) Coronary, Carotid, Illiac, Femoral, and Popitiea Revascularization (Angioplasty/Stent/CABS); n (38, 18, 19, 19, 10) Coronary, Carotid, Illiac, Femoral, and Popitiea Revascularization (Angioplasty/Stent/CABS); n (38, 18, 19, 19, 10) Coronary, Carotid, Illiac, Femoral, and Popitiea Revascularization (Angioplasty/Stent/CABS); n (38, 18, 19, 19 | Acute or Old MI; n (%) | 1,428 (38.8%) | 232 (38.9%) | 0.00 | 713 (24.3%) | 97 (22.5%) | 0.04 | 2,039 (35.0% | 354 (37.6%) | -0.05 | 4,180 (33.6% | 683 (34.7%) | -0.02 |
| Coronary Atheresizerosis, n(%) Coronary Atheresizerosis, n(%) Coronary Atheresizerosis, n(%) Coronary, Carolide, Hillian, Femoria, and Popiliteal Revascularization (Angioplasty/Stert/CABS); n 25(9,8%) 50(8,2%) 50(8,2% | Anxiety; n (%) | 228 (6.2%) | 37 (6.2%) | 0.00 | 125 (4.3%) | 24 (5.6%) | -0.06 | 399 (6.8%) | 58 (6.2%) | 0.02 | 752 (6.0%) | 119 (6.0%) | 0.00 |
| Coronary Carotid, Illiac, Femoral, and Popitreal Revascularization (Angioplasty/Stent/CABC); 1 \$58 (9.7%) 50 (8.4%) 0.05 26 9 (9.2%) 35 (8.1%) 0.04 611 (10.5%) 71 (7.5%) 0.01 327 (12.8%) 0.02 327 (12.8%) 0.02 327 | Atrial Fibrillation; n (%) | 633 (17.2%) | 101 (16.9%) | 0.01 | 387 (13.2%) | 73 (16.9%) | -0.10 | 1,148 (19.7% | 207 (22.0%) | -0.06 | 2,168 (17.4% | 381 (19.3%) | |
| Diabetes with Complications; n (%) | | | 475 (79.6%) | -0.10 | 2,116 (72.0% | 316 (73.3%) | -0.03 | 4,790 (82.2% | 776 (82.5%) | -0.01 | 9,687 (77.8% | 1,567 (79.6% | |
| Diabetes without Complications; n (%) 150 (4.1%) 150 | Coronary, Carotid, Illiac, Femoral, and Popliteal Revascularization (Angioplasty/Stent/CABG); n | 358 (9.7%) | 50 (8.4%) | 0.05 | 269 (9.2%) | 35 (8.1%) | 0.04 | 611 (10.5%) | 71 (7.5%) | 0.10 | 1,238 (9.9%) | 156 (7.9%) | |
| DVT; n(%) | | | | | | | | | | | -, ( | | |
| Edema; n(%) | | | | | | | | | | | | | |
| Erectile dysfunction; n (%) | 7 3 7 | | , , | | | | | | | | | | |
| Foot ulcer; n (%) 90 (2.4%) 23 (3.9%) 9.09 52 (1.8%) 10 (2.3%) 9.04 252 (4.5%) 49 (5.2%) 9.03 40 (3.2%) 82 (4.2%) 9.05 hyperlipidemia; n (%) 9.01 5,288 (3.5%) 3.058 (8.3.9%) 511 (85.6%) 9.05 1,865 (63.5%) 30 (70.1%) 9.01 5,283 (90.6%) 88 (90.2%) 9.02 1,050 (86.2.2 1,671 (84.9%) 9.07 1,000 (1.0.2 1,000 (8.2.2 1,671 (84.9%) 9.07 1,000 (1.0.2 1,000 (8.2.2 1,671 (84.9%) 9.0.0 (8.2.2 1,671 (84.9%) 9.0.0 | | | | | | | | | | | | | |
| Hyperfipidemia; n (%) 3,088 (83.9% \$11 (85.6%) -0.05 1,865 (63.5% 302 (70.1%) -0.14 5,283 (90.6% 858 (91.2%) -0.02 10,236 (82.2 1,671 (84.9%) -0.07 Hypertension; n (%) -0.07 Hypertension; n (%) -0.08 (86.8%) -0.09 1,292 (74.8%) -0.02 1,192 (74.6%) -0.05 1,488 (91.5%) -0.05 1,488 (91.2%) -0.05 1,488 (91.2%) -0.07 1,000 1,00 | | | | | | | | | | | , , | | |
| Hypertension; n (%) 3,188 (86.6%) 522 (87.4%) 4,15%) 5 (0.8%) 5,28 (97.4%) 5,28 (93.1%) 880 (93.5%) 5,428 (93.1%) 880 (93.5%) 5,500 (85.7%) 880 (85.7%) 5,500 (85.7%) 880 (85.7% | | ( ' ' ' | | | - ( / | | | | | | | | |
| Intracranial or Retroperitoneal Hemorrhage; n (%) 54 (1.5%) 50 (1.5%) 50 (1.5%) 50 (1.5%) 50 (1.5%) 50 (1.2%) -0.05 50 (1.2%) -0.04 50 (1.5%) -0.05 50 (1.5%) -0.05 50 (1.5%) -0.05 50 (1.5%) -0.05 50 (1.5%) -0.05 50 (1.5%) -0.06 50 (1.5%) -0.06 50 (1.5%) -0.07 50 (1.5%) -0. | | | | | | | | | | | | | <u> </u> |
| Ischemic Heart Disease; n (%) 3,026 (82.2%) 504 (84.4%) -0.06 2,250 (76.6%) 333 (77.3%) -0.02 5,000 (85.8%) 806 (85.7%) -0.00 10,276 (82.6] 1,643 (83.4%) -0.02 1,510 (25.9%) 232 (24.7%) -0.03 2,551 (21.3%) 430 (21.8%) -0.01 4,41 (1.8%) -0.04 4,11 (1.5%) -0.04 4, | | | | | , , | | | | | | | | <u> </u> |
| Ischemic Stroke; n (%) 644 (17.5%) 19 (19.9%) -0.06 497 (16.9%) 79 (18.3%) -0.04 1,510 (25.9%) 232 (24.7%) 0.03 2,651 (21.3%) 430 (21.8%) -0.01 | | | | | | | | | | | | | |
| Major Trauma; n (%) | | | | | | | | | | | | | |
| Obesity; n (%) 524 (14.2%) 68 (11.4%) 0.08 (25.86%) 47 (10.9%) -0.08 (97.61.7%) 164 (17.4%) -0.02 (1,752 (14.1%) 279 (14.2%) 0.00 Other Disorders of Thyroid Gland; n (%) 112 (3.0%) 18 (3.0%) 0.00 (69 (2.3%)) 13 (3.0%) -0.04 (26 (4.5%)) 38 (4.0%) 0.02 (443 (3.6%)) 69 (3.5%) 0.01 Overweight; n (%) 294 (8.0%) 46 (7.7%) 0.01 (83 (3.8%)) 13 (3.0%) -0.01 (20 (8.6%)) 42 (4.5%) -0.05 (885 (4.7%)) -0.05 (885 (4.7%)) 0.02 (97 (1.6%)) -0.02 Peripheral Vascular Disease; n (%) 1,234 (33.5%) 205 (34.3%) -0.02 (75 (24.0%)) 117 (27.1%) -0.07 (1,798 (30.8%) 277 (29.4%) 0.03 (3,737 (30.0%) 599 (3.4%) -0.01 Systemic Embolism; n (%) 490 (13.3%) 83 (13.9%) -0.02 (276 (9.4%)) 37 (8.6%) 0.03 (769 (13.2%)) 115 (12.2%) 0.03 (1,535 (12.3%) 295 (11.9%) 0.01 Systemic Embolism; n (%) 60 (1.6%) 11 (1.8%) -0.02 (49 (1.7%)) 10 (2.3%) -0.04 N/A N/A N/A N/A N/A Abnormal liver function; n (%) 333 (9.0%) 55 (9.2%) -0.01 (189 (6.4%)) 28 (6.5%) | , , , | . , | | | | | | | , , | | | | |
| Other Disorders of Thyroid Gland; n (%) 112 (3.0%) 18 (3.0%) 0.00 69 (2.3%) 13 (3.0%) 0.01 83 (2.8%) 13 (3.0%) 0.01 208 (3.6%) 12 (4.5%) 18 (4.0%) 0.02 443 (3.6%) 69 (3.5%) 0.01 208 (3.6%) 10 (1.5%) 0.02 49 (1.5%) 10 (1.5%) 0.02 18 (2.8%) 10 (1.5%) 0.01 208 (3.6%) 10 (1.7%) 0.01 39 (1.3%) 10 (1.7%) 0.02 49 (1.3%) 10 (1.7%) 1 | | | | | | | | | | | | | |
| Overweight; n (%) 294 (8.0%) 46 (7.7%) 0.01 83 (2.8%) 13 (3.0%) -0.01 208 (3.6%) 42 (4.5%) -0.05 585 (4.7%) 10 (1.5%) -0.02 197 (1.6%) 10 (1.7%) -0.01 39 (1.3%) 20.5%) 0.08 99 (1.7%) 14 (1.5%) 0.02 197 (1.6%) 10 (5.1%) 0.02 197 (1.6%) 10 (5.1%) 0.03 1,234 (33.5%) 205 (34.3%) -0.02 705 (24.0%) 17 (27.1%) -0.07 1,798 (30.8%) 277 (29.4%) 0.03 3,737 (30.0%) 599 (30.4%) -0.01 254 (3.3%) 0.02 197 (1.6%) 26 (1.3%) 0.03 1,535 (12.3%) 255 (1.9%) 0.01 Systemic Embolism; n (%) 0.02 276 (9.4%) 37 (8.6%) 0.03 3769 (13.2%) 15 (1.2%) 0.03 1,535 (12.3%) 235 (11.9%) 0.01 Systemic Embolism; n (%) 0.02 276 (9.4%) 17 (27.1%) 0.07 1,798 (30.8%) 17 (9.1%) 15 (12.2%) 0.03 1,535 (12.3%) 235 (11.9%) 0.01 15 (12.5%) 0.03 1,535 (12.3%) 25 (1.9%) 0.01 15 (12.5%) 0.03 1,535 (12.3%) 25 (1.9%) 0.01 15 (12.5%) 0.03 1,535 (12.3%) 25 (1.9%) 0.01 15 (12.5%) 0.03 1,535 (12.3%) 25 (1.9%) 0.01 15 (12.5%) 0.03 1,535 (12.3%) 25 (1.9%) 0.01 15 (12.5%) 0.03 1,535 (12.3%) 0.03 1,535 | | - ( - / | | | | ( / | | ( / | | | | | |
| PE; n (%) 59 (1.6%) 10 (1.7%) -0.01 39 (1.3%) 2 (0.5%) 0.08 99 (1.7%) 14 (1.5%) 0.02 197 (1.6%) 26 (1.3%) 0.03 Peripheral Vascular Disease; n (%) 1,234 (33.5%) 205 (34.3%) -0.02 705 (24.0%) 117 (27.1%) -0.07 1,798 (30.8%) 277 (29.4%) 0.03 3,737 (30.0%) 599 (30.4%) -0.01 Stable Angina; n (%) 490 (13.3%) 83 (13.9%) -0.02 276 (9.4%) 37 (8.6%) 0.03 76 (91.2%) 115 (12.2%) 0.03 1,535 (12.3%) 235 (11.9%) -0.01 Systemic Embolism; n (%) 60 (1.6%) 11 (1.8%) -0.02 49 (1.7%) 10 (2.3%) -0.04 N/A | | | | | | | | | | | | | |
| Peripheral Vascular Disease; n (%) 1,234 (33.5% 205 (34.3%) -0.02 705 (24.0%) 17 (27.1%) -0.07 1,798 (30.8% 277 (29.4%) 0.03 3,737 (30.0% 599 (30.4%) -0.01 Stable Angina; n (%) 490 (13.3%) 83 (13.9%) -0.02 276 (9.4%) 37 (8.6%) 0.03 769 (13.2%) 115 (12.2%) 0.03 1,535 (12.3% 235 (11.9%) 0.01 Systemic Embolism; n (%) 60 (1.6%) 11 (1.8%) -0.02 49 (1.7%) 10 (2.3%) -0.04 N/A | | | , , | | . , | | | | | | | | |
| Stable Angina; n (%) | | | | | | | | | | | | | |
| Systemic Embolism; n (%) 60 (1.6%) 11 (1.8%) -0.02 49 (1.7%) 10 (2.3%) -0.04 N/A | | | | | | | | | | | | | |
| TIA; n (%) 90 (2.4%) 22 (3.7%) -0.08 63 (2.1%) 10 (2.3%) -0.01 266 (4.6%) 36 (3.8%) 0.04 419 (3.4%) 68 (3.5%) -0.01<br>General Health/Mortality Prognosticators Abnormal liver function; n (%) 333 (9.0%) 55 (9.2%) -0.01 189 (6.4%) 28 (6.5%) 0.00 574 (9.8%) 97 (10.3%) -0.02 1,096 (8.8%) 180 (9.1%) -0.01 Alcohol Abuse/Dependence; n (%) -0.01 108 (1.9%) 19 (2.0%) -0.01 108 (1.9%) 19 (2.0%) -0.01 213 (1.7%) 41 (2.1%) -0.03 Asthma; n (%) -0.04 40 (2.8%) 157 (26.3%) -0.08 492 (16.7%) 72 (16.7%) -0.01 108 (1.9%) 19 (2.0%) -0.01 213 (1.7%) 515 (2.2%) -0.01 Asthma; n (%) -0.02 1,096 (8.8%) 180 (9.1%) -0.03 -0.03 Asthma; n (%) -0.03 1,000 1 | 5 , t , | | | | | | | . , | | | , , | | |
| General Health/Mortality Prognosticators 333 (9.0%) 55 (9.2%) -0.01 189 (6.4%) 28 (6.5%) 0.00 574 (9.8%) 97 (10.3%) -0.02 1,096 (8.8%) 180 (9.1%) -0.01 Alcohol Abuse/Dependence; n (%) Alcohol Abuse/Dependence; n (%) 72 (2.0%) 17 (2.8%) -0.05 33 (1.1%) 5 (1.2%) -0.01 108 (1.9%) 19 (2.0%) -0.01 213 (1.7%) 41 (2.1%) -0.03 Anemias (Sickle-Cell, G6PD Deficiency, Nutrient Deficiency); n (%) 840 (22.8%) 157 (26.3%) -0.08 492 (16.7%) 72 (16.7%) 0.00 1 (19 (1.9%) 19 (2.0%) -0.01 213 (1.7%) 41 (2.1%) -0.03 Anemias (10 (1.9%) 19 (2.0%) -0.01 213 (1.7%) 41 (2.1%) -0.03 Anemias (10 (1.9%) 19 (2.0%) -0.01 213 (1.7%) 41 (2.1%) -0.03 Anemias (10 (1.9%) 19 (2.0%) -0.01 213 (1.7%) 41 (2.1%) -0.03 Anemias (10 (1.9%) 19 (2.0%) -0.01 213 (1.7%) 41 (2.1%) -0.03 Anemias (10 (1.9%) -0.01 213 (1.7%) 41 (2.1%) -0.03 Anemias (10 (1.9%) -0.01 213 (1.7%) 41 (2.1%) -0.03 Anemias (10 (1.9%) -0.01 213 (1.7%) 41 (2.1%) -0.03 Anemias (10 (1.9%) -0.01 213 (1.7%) -0.01 213 (1.7%) -0.01 213 (1.7%) -0.01 213 (1.7%) -0.01 213 (1.7%) | | | | | | | | | | | | | |
| Abnormal liver function; n (%) 333 (9.0%) 55 (9.2%) -0.01 189 (6.4%) 28 (6.5%) 0.00 574 (9.8%) 97 (10.3%) -0.02 1,096 (8.8%) 180 (9.1%) -0.01 Alcohol Abuse/Dependence; n (%) 72 (2.0%) 17 (2.8%) -0.05 33 (1.1%) 5 (1.2%) -0.01 108 (1.9%) 19 (2.0%) -0.01 213 (1.7%) 41 (2.1%) -0.03 Anemias (Sickle-Cell, G6PD Deficiency, Nutrient Deficiency); n (%) 840 (22.8%) 157 (26.3%) -0.08 492 (16.7%) 72 (16.7%) -0.00 1,970 (33.8%) 286 (30.4%) -0.07 3,302 (26.5%) 15 (62.2%) -0.01 Asthma; n (%) -0.01 (108 (1.9%) 150 (4.1%) 22 (3.7%) -0.02 106 (3.6%) 22 (5.1%) -0.07 351 (6.0%) 58 (6.2%) -0.01 607 (4.9%) 102 (5.2%) -0.01 COPD; n (%) -0.01 (108 (1.9%) 150 (4.1%) 22 (3.7%) -0.01 (108 (1.9%) 150 (4.1%) 22 (3.7%) -0.01 (108 (1.9%) 150 (4.1%) 22 (3.7%) -0.01 (108 (1.9%) 150 (4.1%) 150 | | () | (5 /5) | 2.00 | (/-) | (2.5/0) | 5.01 | (,) | (5.575) | 3.04 | 5 (5. 1,0) | 23 (3.370) | 0.01 |
| Alcohol Abuse/Dependence; n (%) 72 (2.0%) 17 (2.8%) -0.05 33 (1.1%) 5 (1.2%) -0.01 108 (1.9%) 19 (2.0%) -0.01 213 (1.7%) 41 (2.1%) -0.03 Anemias (Sickle-Cell, G6PD Deficiency, Nutrient Deficiency); n (%) 840 (22.8%) 157 (26.3%) -0.08 492 (16.7%) 72 (16.7%) 0.00 1,970 (33.8%) 286 (30.4%) 0.07 3,302 (26.5%) 515 (26.2%) 0.01 Asthma; n (%) 150 (4.1%) 22 (3.7%) 0.02 106 (3.6%) 22 (5.1%) -0.07 351 (6.0%) 58 (6.2%) -0.01 607 (4.9%) 102 (5.2%) -0.01 COPD; n (%) 859 (23.3%) 137 (22.9%) 0.01 502 (17.1%) 79 (18.3%) -0.03 1,421 (24.4%) 223 (23.7%) 0.02 2,782 (22.3%) 439 (22.3%) 0.00 | | 333 (9.0%) | 55 (9.2%) | -0.01 | 189 (6.4%) | 28 (6.5%) | 0.00 | 574 (9.8%) | 97 (10.3%) | -0.02 | 1.096 (8.8%) | 180 (9.1%) | -0.01 |
| Anemias (Sickle-Cell, G6PD Deficiency, Nutrient Deficiency); n (%) 840 (22.8%) 157 (26.3%) -0.08 492 (16.7%) 72 (16.7%) 0.00 1,970 (33.8% 286 (30.4%) 0.07 3,302 (26.5% 515 (26.2%) 0.01 25.2%) -0.01 25.2% -0. | | | , , | | | | | | | | | | |
| Ashma; n (%) | | | | | . , | | | | | | | | |
| COPD, n (%) 859 (23.3%) 137 (22.9%) 0.01 502 (17.1%) 79 (18.3%) -0.03 1,421 (24.4% 223 (23.7%) 0.02 2,782 (22.3% 439 (22.3%) 0.00 | | | | | | | | | | | | | |
| | Delirium; n (%) | | | | | | | | | | | | |

# Table 1 Unmatched

| Dementia; n (%) | 101 (2.7%) | 18 (3.0%) | -0.02 | 56 (1.9%) | 10 (2.3%) | -0.03 | 222 (3.8%) | 31 (3.3%) | 0.03 | 3 379 (3.0%) | 59 (3.0%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Depression ; n (%) | 318 (8.6%) | 48 (8.0%) | 0.02 | 157 (5.3%) | 25 (5.8%) | -0.02 | 561 (9.6%) | 77 (8.2%) | 0.0 | 5 1,036 (8.3%) | 150 (7.6%) | 0.03 |
| Falls; n (%) | 229 (6.2%) | 42 (7.0%) | -0.03 | 68 (2.3%) | 13 (3.0%) | -0.04 | 351 (6.0%) | 72 (7.7%) | -0.0 | 7 648 (5.2%) | 127 (6.4%) | -0.05 |
| Fractures; n (%) | 226 (6.1%) | 32 (5.4%) | 0.03 | 147 (5.0%) | 22 (5.1%) | 0.00 | 341 (5.9%) | 47 (5.0%) | 0.04 | 4 714 (5.7%) | 101 (5.1%) | 0.03 |
| HIV/AIDS; n (%) | 6 (0.2%) | 2 (0.3%) | -0.02 | 1 (0.0%) | 0 (0.0%) | | N/A | N/A | N/A | N/A | N/A | N/A |
| Organ Transplant; n (%) | 16 (0.4%) | 5 (0.8%) | -0.05 | 20 (0.7%) | 4 (0.9%) | -0.02 | | N/A | N/A | N/A | N/A | N/A |
| Osteoporosis; n (%) | 201 (5.5%) | 27 (4.5%) | 0.05 | | 14 (3.2%) | | | 56 (6.0%) | | 3 734 (5.9%) | 97 (4.9%) | 0.04 |
| Peptic Ulcer Disease; n (%) | 892 (24.2%) | 154 (25.8%) | | 437 (14.9%) | 80 (18.6%) | | 1,593 (27.3% | | | 2,922 (23.5% | | -0.04 |
| Pneumonia; n (%) | 72 (2.0%) | 17 (2.8%) | | 134 (4.6%) | 17 (3.9%) | | | 19 (2.0%) | -0.03 | | 53 (2.7%) | -0.04 |
| Renal Failure; n (%) | 775 (21.1%) | 142 (23.8%) | -0.05 | | | | 1,467 (25.2% | | | 4 2,635 (21.2% | | -0.04 |
| Renal Failure (CKD Stage 4 or higher); n (%) | 128 (3.5%) | 20 (3.4%) | 0.01 | 95 (3.2%) | 12 (2.8%) | | | 50 (5.3%) | 0.00 | | 82 (4.2%) | 0.00 |
| Sleep Apnea; n (%) | 432 (11.7%) | 57 (9.5%) | 0.07 | 317 (10.8%) | 44 (10.2%) | | | 109 (11.6%) | | 3 1,490 (12.0% | | 0.04 |
| Sleep Disorder; n (%) | 295 (8.0%) | 29 (4.9%) | 0.13 | 307 (10.4%) | 39 (9.0%) | 0.05 | | | 0.00 | _ ` ` ` | | 0.07 |
| Smoking; n (%) | 1,015 (27.6% | 194 (32.5%) | -0.11 | 352 (12.0%) | 71 (16.5%) | -0.13 | 1,758 (30.2% | 296 (31.5%) | -0.03 | 3,125 (25.1% | 561 (28.5%) | -0.08 |
| Frailty Score: Empirical Version 365 days (ICD-9 and ICD-10) v2 | | | | | | | | | | | | |
| mean (sd) | 0.17 (0.05) | 0.17 (0.05) | | 0.16 (0.05) | 0.16 (0.05) | | | 0.19 (0.06) | | 7 0.18 (0.05) | 0.18 (0.06) | 0.00 |
| median [IQR] | 0.16 [0.13, 0. | 0.16 [0.13, 0. | 0.00 | 0.15 [0.13, 0 | . 0.15 [0.13, 0. | 0.00 | 0.19 [0.16, 0. | 0.18 [0.15, 0. | 0.1 | 7 0.17 (0.06) | 0.17 (0.06) | 0.00 |
| Healthcare utilization | | | | | | | | | | | | |
| Any hospitalization; n (%) | 905 (24.6%) | 155 (26.0%) | -0.03 | 786 (26.8%) | 95 (22.0%) | 0.11 | 1,691 (29.0% | 250 (26.6%) | 0.0 | 3,382 (27.2% | | 0.04 |
| Bone mineral density; n (%) | 162 (4.4%) | 23 (3.9%) | 0.03 | 78 (2.7%) | 10 (2.3%) | 0.03 | 245 (4.2%) | 43 (4.6%) | -0.02 | 2 485 (3.9%) | 76 (3.9%) | 0.00 |
| BUN tests; n (%) | 502 (13.6%) | 89 (14.9%) | | 281 (9.6%) | 48 (11.1%) | | 1,151 (19.7% | | | 1,934 (15.5% | | -0.02 |
| Cardiologist visit | 1 | | | · · · · · · · | 1 | | | , · · · · · | | 1 | | |
| 0 | 1.492 (40.5% | 205 (34.3%) | 0.13 | 1,317 (44.8% | 193 (44.8%) | 0.00 | 1,338 (23.0% | 195 (20.7%) | 0.00 | 5 4,147 (33.3% | 593 (30.1%) | 0.07 |
| 1-2 | | 175 (29.3%) | | 744 (25.3%) | | | 1,920 (32.9% | | | 3 3,765 (30.2% | | -0.02 |
| 3-5 | 665 (18.1%) | 146 (24.5%) | -0.16 | | | | 1,567 (26.9% | | | 2,768 (22.2% | | -0.05 |
| >=6 | 423 (11.5%) | 71 (11.9%) | -0.10 | 341 (11.6%) | | | 1,004 (17.2% | | -0.03 | | 285 (14.5%) | -0.03 |
| | 412 (11.2%) | 69 (11.6%) | -0.01 | 330 (11.2%) | 43 (10.0%) | | , , | 109 (11.6%) | -0.03 | _ ` ` ` | 221 (11.2%) | -0.01 |
| Colonoscopy; n (%) | | | | | | | | | -0.03 | | | 0.00 |
| Endocrinologist Visit; n (%) | 178 (4.8%) | 20 (3.4%) | 0.07 | 83 (2.8%) | 15 (3.5%) | | | 93 (9.9%) | | | 128 (6.5%) | |
| Fecal occult blood (FOB) test; n (%) | 300 (8.1%) | 52 (8.7%) | -0.02 | 127 (4.3%) | 20 (4.6%) | | | 64 (6.8%) | | 828 (6.7%) | 136 (6.9%) | -0.01 |
| Flu vaccine; n (%) | | 218 (36.5%) | -0.01 | . , | | | 3,495 (60.0% | | | 2 5,416 (43.5% | | -0.06 |
| Glucose test strips; n (%) | 86 (2.3%) | 14 (2.3%) | 0.00 | 45 (1.5%) | 8 (1.9%) | | 357 (6.1%) | 63 (6.7%) | | 2 488 (3.9%) | 85 (4.3%) | -0.02 |
| Glucose tests; n (%) | 578 (15.7%) | 101 (16.9%) | -0.03 | | 59 (13.7%) | | 1,837 (31.5% | | | 5 2,751 (22.1% | | 0.00 |
| HbA1c tests ; n (%) | 1,554 (42.2% | 280 (46.9%) | -0.09 | 570 (19.4%) | 97 (22.5%) | -0.08 | 4,510 (77.4% | 724 (76.9%) | 0.03 | 1 6,634 (53.3% | 1,101 (55.9% | -0.05 |
| Imaging/Diagnostics Used in Prostate Cancer | | | | | | | | | | | | |
| 0 | 1,717 (46.6% | 197 (33.0%) | 0.28 | 1,366 (46.5% | 132 (30.6%) | 0.33 | 2,879 (49.4% | 355 (37.7%) | 0.24 | 4 5,962 (47.9% | 684 (34.7%) | 0.27 |
| 1-3 | 1,620 (44.0% | 323 (54.1%) | -0.20 | 1,243 (42.3% | 217 (50.3%) | -0.16 | 2,248 (38.6% | 438 (46.5%) | -0.16 | 5,111 (41.1% | 978 (49.7%) | -0.17 |
| >=4 | 344 (9.3%) | 77 (12.9%) | -0.11 | 329 (11.2%) | 82 (19.0%) | -0.22 | 702 (12.0%) | 148 (15.7%) | -0.13 | 1 1,375 (11.0% | 307 (15.6%) | -0.14 |
| Internal Medicine/Family Medicine Visits; n (%) | 3,489 (94.8% | 568 (95.1%) | -0.01 | 2,513 (85.5% | 377 (87.5%) | -0.06 | 5,219 (89.5% | 838 (89.1%) | 0.0 | 1 11,221 (90.1 | 1,783 (90.6% | -0.02 |
| Lipid tests; n (%) | 2,689 (73.1% | 439 (73.5%) | -0.01 | 1,011 (34.4% | 152 (35.3%) | -0.02 | 5,013 (86.0% | 789 (83.8%) | 0.0 | 8,713 (70.0% | 1,380 (70.1% | 0.00 |
| Microalbuminuria tests; n (%) | 921 (25.0%) | 150 (25.1%) | 0.00 | 404 (13.8%) | 72 (16.7%) | -0.08 | 2,428 (41.7% | 425 (45.2%) | | 7 3,753 (30.1% | | -0.06 |
| Number of different/distinct medication prescriptions | , , , , , | , , , , | | , , , , , | , , , , | | , , , , , , | , , , , | | , | ( / | |
| mean (sd) | 8.01 (6.17) | 8.27 (6.02) | -0.04 | 10 22 (5 52) | 10.55 (5.10) | -0.06 | 11.92 (5.24) | 11 69 (4 90) | 0.01 | 5 10.36 (5.60) | 10 40 (5 31) | -0.01 |
| median [IQR] | | 8.00 [4.00, 12 | | | 3 10.00 [7.00, | | 11.00 [8.00, 1 | | | 9.64 (6.20) | | -0.04 |
| Office Visits (outpatient setting only) | 0.00 (0.00) 11 | 0.00 (1.00, 1. | 0.00 | 3.00 (0.00, 1 | 10.00 (7.00) | 0.13 | 11.00 (0.00) | 11.00 (0.00) | 0.00 | 3.0. (0.20) | 3.07 (3.32) | 0.0 |
| mean (sd) | 12 49 (6 90) | 12.44 (6.38) | 0.01 | 12 21 /7 02\ | 12.46 (6.32) | 0.02 | 14.62 (7.67) | 14 20 (6 05) | 0.01 | 5 13.44 (7.27) | 12 22 /6 65\ | 0.02 |
| | | 11.00 [8.00, | | | 111.00 [8.00, | | 13.00 [9.00, 1 | | | 0 11.94 (8.02) | | 0.02 |
| median [IQR] | 11.00 [8.00, 1 | 11.00 [8.00, | 15.00] | 11.00 [8.00, | 111.00 [8.00, | 0.00 | 13.00 [9.00, 1 | 13.00 [9.00, . | 0.00 | 7 11.94 (8.02) | 11.90 (7.38) | 0.00 |
| Oncology Specialist Visit | 2 574 /60 00/ | 1 400 (50 50() | 0.00 | 2 550 (00 00 | ( 200 (00 50() | 0.04 | 2 246 (55 70) | 552 (50 70() | 0.00 | | 4 254 (60 60) | |
| 0 | 2,571 (69.8% | | | 2,668 (90.8% | | | 3,246 (55.7% | | | 8,485 (68.2% | | -0.01 |
| 1-5 | | 77 (12.9%) | | 112 (3.8%) | 16 (3.7%) | | 1,059 (18.2% | | | 1,626 (13.1% | | -0.03 |
| >=6 | 655 (17.8%) | 111 (18.6%) | | . , | 25 (5.8%) | -0.02 | , , | | | 2,337 (18.8% | | 0.04 |
| Pneumonia vaccine; n (%) | 958 (26.0%) | 183 (30.7%) | -0.10 | 276 (9.4%) | 49 (11.4%) | -0.07 | 1,445 (24.8% | 281 (29.9%) | -0.1 | 1 2,679 (21.5% | 513 (26.1%) | -0.11 |
| Prostate cancer prognosticators | | | | | | | | | | | | |
| Radiation Therapies Used in Prostate Cancer; n (%) | 18 (0.5%) | 1 (0.2%) | 0.05 | 7 (0.2%) | 0 (0.0%) | 0.06 | N/A | N/A | N/A | N/A | N/A | N/A |
| PSA Test | | | | | | | | | | | | |
| mean (sd) | 2.42 (1.78) | 2.40 (1.74) | 0.01 | 1.19 (3.39) | 1.00 (1.51) | 0.12 | 2.59 (1.58) | 2.41 (1.43) | 0.12 | 2 2.21 (2.20) | 2.10 (1.55) | 0.06 |
| median [IQR] | 2.00 [1.00, 3. | 2.00 [1.00, 3. | | | 0.00 [0.00, 2. | | 2.00 [2.00, 3. | | | 3 1.53 (2.74) | 1.56 (1.73) | -0.01 |
| Prostatectomy; n (%) | 146 (4.0%) | 18 (3.0%) | | 117 (4.0%) | 11 (2.6%) | | 132 (2.3%) | 22 (2.3%) | | 395 (3.2%) | 51 (2.6%) | 0.04 |
| Prostate exam for DRE | . , | - ,,- | 2.33 | ,/ | , -,-, | 2.30 | - ,,-, | , -,-, | 1.0 | (2.2.7.7) | , -,-, | 5.0 |
| mean (sd) | 1.19 (3.27) | 1.18 (2.90) | 0.00 | 0.31 (1.48) | 0.31 (1.42) | 0 17 | 0.38 (0.81) | 0.42 (0.82) | -0.0 | 5 | | |
| median [IQR] | | 0.00 [0.00, 0. | | | . 0.00 [0.00, 0. | | 0.00 [0.00, 0. | | 0.00 | | l | <b>-</b> |
| Prostate Cancer Comorbidity Index (PCCI) | J.00 [0.00, 0. | 0.00 [0.00, 0. | 0.00 | 0.00 [0.00, 0 | . 5.55 [0.55, 0. | 0.17 | 0.00 [0.00, 0. | 0.00 [0.00, 1. | 0.00 | 1 | t | <del> </del> |
| | 25 65 16 071 | 26 60 16 241 | 0.17 | 22 24 (4 00) | 24 65 /5 27\ | 0.03 | 26 26 16 001 | 26 00 /6 27\ | 0.14 | 25 44 (5 70) | 26 20 16 16\ | -0.16 |
| mean (sd) | | 36.68 (6.34) | | 33.34 (4.90) | | | 36.36 (6.00) | | | 35.44 (5.78) | | |
| median [IQR] | 35.00 [31.00, | 36.00 [32.00 | , 0.00 | 33.00 [30.00 | , 34.00 [30.00 | , -0.02 | 35.00 [32.00, | 30.00 [33.00] | -0.16 | 34.53 (6.24) | 35.56 (6.74) | -0.16 |
| Medications | | I | | | | | | | | | | |
| ACE inhibitors; n (%) | 1,263 (34.3% | 190 (31.8%) | 0.05 | 1,161 (39.5% | 181 (42.0%) | -0.05 | 2,704 (46.4% | 461 (49.0%) | -0.0 | 5,128 (41.2% | 832 (42.3%) | -0.02 |

# Table 1 Unmatched

| Anti-arrhythmics; n (%) | 54 (1.5%) | 12 (2.0%) | -0.04 5 | 5 (1.9%) | 5 (1.2%) | 0.06 | 136 (2.3%) | 20 (2.1%) | | 0.01 | 245 (2.0%) | 37 (1.9%) | | 0.01 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Anti-diabetic Drugs; n (%) | 747 (20.3%) | 131 (21.9%) | -0.04 | 52 (25.6%) | 118 (27.4%) | -0.04 | 3,789 (65.09 | 582 (61.8%) | | 0.07 | 5,288 (42.5% | 831 (42.2%) | | 0.01 |
| Chemotherapies Used in Prostate Cancer; n (%) | 18 (0.5%) | 1 (0.2%) | 0.05 1 | .0 (0.3%) | 0 (0.0%) | 0.08 | N/A | N/A | N/A | | N/A | N/A | N/A | |
| Metformin; n (%) | 486 (13.2%) | 87 (14.6%) | -0.04 | 88 (13.2%) | 68 (15.8%) | -0.07 | 2,144 (36.89 | 346 (36.8%) | | 0.00 | 3,018 (24.2% | 501 (25.4%) | | -0.03 |
| Use of anticonvulsants; n (%) | 354 (9.6%) | 52 (8.7%) | 0.03 2 | 93 (10.0%) | 44 (10.2%) | -0.01 | 901 (15.5%) | 138 (14.7%) | | 0.02 | 1,548 (12.4% | 234 (11.9%) | | 0.02 |
| Use of antidepressants; n (%) | 426 (11.6%) | 70 (11.7%) | 0.00 3 | 79 (12.9%) | 58 (13.5%) | -0.02 | 1,015 (17.49 | 6 144 (15.3%) | | 0.06 | 1,820 (14.6% | 272 (13.8%) | | 0.02 |
| Use of Antiparkinsonian Meds; n (%) | 51 (1.4%) | 13 (2.2%) | -0.06 | 9 (2.3%) | 7 (1.6%) | 0.05 | 207 (3.6%) | 18 (1.9%) | | 0.10 | 327 (2.6%) | 38 (1.9%) | | 0.05 |
| Use of antiplatelet agents; n (%) | 985 (26.8%) | 161 (27.0%) | 0.00 1 | ,135 (38.6% | 162 (37.6%) | 0.02 | 2,276 (39.09 | 356 (37.8%) | | 0.02 | 4,396 (35.3% | 679 (34.5%) | | 0.02 |
| Use of antipsychotics; n (%) | 25 (0.7%) | 7 (1.2%) | -0.05 | 5 (1.2%) | 8 (1.9%) | -0.06 | N/A | N/A | N/A | | N/A | N/A | N/A | |
| Use of anxiolytics/hypnotics; n (%) | 137 (3.7%) | 25 (4.2%) | -0.03 1 | 76 (6.0%) | 25 (5.8%) | 0.01 | 428 (7.3%) | 62 (6.6%) | | | | 112 (5.7%) | | 0.01 |
| Use of ARBs; n (%) | 573 (15.6%) | 100 (16.8%) | -0.03 € | 27 (21.3%) | 88 (20.4%) | 0.02 | 1,403 (24.19 | 230 (24.4%) | | -0.01 | 2,603 (20.9% | 418 (21.2%) | | -0.01 |
| Use of Benzos; n (%) | 355 (9.6%) | 60 (10.1%) | -0.02 4 | 09 (13.9%) | 45 (10.4%) | 0.11 | 594 (10.2%) | 108 (11.5%) | | -0.04 | 1,358 (10.9% | 213 (10.8%) | | 0.00 |
| Use of beta blockers; n (%) | 1,806 (49.1% | 305 (51.1%) | -0.04 1 | ,879 (64.0% | 286 (66.4%) | -0.05 | 3,987 (68.49 | 689 (73.2%) | | -0.11 | 7,672 (61.6% | 1,280 (65.0% | 6 | -0.07 |
| Use of bisphosphonate; n (%) | 105 (2.9%) | 9 (1.5%) | 0.10 8 | 2 (2.8%) | 5 (1.2%) | 0.11 | 175 (3.0%) | 18 (1.9%) | | 0.07 | 362 (2.9%) | 32 (1.6%) | | 0.09 |
| Use of calcium channel blockers; n (%) | 837 (22.7%) | 154 (25.8%) | -0.07 | 89 (30.3%) | 113 (26.2%) | 0.09 | 1,955 (33.5% | 6 294 (31.2%) | | 0.05 | 3,681 (29.6% | 561 (28.5%) | | 0.02 |
| Use of COPD/asthma meds; n (%) | 468 (12.7%) | 82 (13.7%) | -0.03 5 | 13 (17.5%) | 89 (20.6%) | -0.08 | 1,128 (19.49 | 6 166 (17.6%) | | 0.05 | 2,109 (16.9% | 337 (17.1%) | | -0.01 |
| Use of Dementia Meds; n (%) | 30 (0.8%) | 10 (1.7%) | -0.08 | 3 (2.1%) | 8 (1.9%) | 0.01 | 153 (2.6%) | 19 (2.0%) | | 0.04 | 246 (2.0%) | 37 (1.9%) | | 0.01 |
| Use of digoxin; n (%) | 53 (1.4%) | 12 (2.0%) | -0.05 | 3 (3.2%) | 12 (2.8%) | 0.02 | 211 (3.6%) | 43 (4.6%) | | -0.05 | 357 (2.9%) | 67 (3.4%) | | -0.03 |
| Use of heparin and other low-molecular weight heparins; n (%) | 40 (1.1%) | 8 (1.3%) | -0.02 € | 2 (2.1%) | 7 (1.6%) | 0.04 | 107 (1.8%) | 25 (2.7%) | | -0.06 | 209 (1.7%) | 40 (2.0%) | | -0.02 |
| Use of Insulin; n (%) | 214 (5.8%) | 34 (5.7%) | 0.00 2 | 23 (7.6%) | 34 (7.9%) | -0.01 | 1,154 (19.89 | 6 186 (19.8%) | | 0.00 | 1,591 (12.8% | 254 (12.9%) | | 0.00 |
| Use of Lithium; n (%) | 6 (0.2%) | 0 (0.0%) | 0.06 2 | (0.1%) | 0 (0.0%) | 0.04 | N/A | N/A | N/A | | N/A | N/A | N/A | |
| Use of Loop Diuretics; n (%) | 338 (9.2%) | 59 (9.9%) | -0.02 3 | 95 (13.4%) | 61 (14.2%) | -0.02 | 1,199 (20.69 | 6 197 (20.9%) | | -0.01 | 1,932 (15.5% | 317 (16.1%) | | -0.02 |
| Use of nitrates; n (%) | 524 (14.2%) | 75 (12.6%) | 0.05 | 30 (21.4%) | 82 (19.0%) | 0.06 | 1,348 (23.19 | 6 205 (21.8%) | | 0.03 | 2,502 (20.1% | 362 (18.4%) | | 0.04 |
| Use of NSAIDs; n (%) | 405 (11.0%) | 74 (12.4%) | -0.04 4 | 02 (13.7%) | 57 (13.2%) | 0.01 | 1,015 (17.49 | 6 132 (14.0%) | | 0.09 | 1,822 (14.6% | 263 (13.4%) | | 0.03 |
| Use of opioids; n (%) | 1,034 (28.1% | 173 (29.0%) | -0.02 1 | ,087 (37.0% | 171 (39.7%) | -0.06 | 2,338 (40.19 | 369 (39.2%) | | 0.02 | 4,459 (35.8% | 713 (36.2%) | | -0.01 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, Apixaban, Warfarin); n (%) | 326 (8.9%) | 52 (8.7%) | 0.01 3 | 50 (11.9%) | 53 (12.3%) | -0.01 | 822 (14.1%) | 147 (15.6%) | | -0.04 | 1,498 (12.0% | 252 (12.8%) | | -0.02 |
| Use of oral corticosteroids; n (%) | 700 (19.0%) | 134 (22.4%) | -0.08 7 | 10 (24.2%) | 103 (23.9%) | 0.01 | 1,538 (26.49 | 252 (26.8%) | | -0.01 | 2,948 (23.7% | 489 (24.8%) | | -0.03 |
| Use of other antiplatelet agents; n (%) | 33 (0.9%) | 8 (1.3%) | -0.04 5 | 0 (1.7%) | 3 (0.7%) | 0.09 | N/A | N/A | N/A | | N/A | N/A | N/A | |
| Use of other diuretics; n (%) | 100 (2.7%) | 16 (2.7%) | 0.00 1 | .22 (4.2%) | 22 (5.1%) | | | 52 (5.5%) | | -0.02 | 511 (4.1%) | 90 (4.6%) | | -0.02 |
| Use of other hypertension drugs; n (%) | 274 (7.4%) | 49 (8.2%) | -0.03 2 | 66 (9.1%) | 32 (7.4%) | 0.06 | 661 (11.3%) | 91 (9.7%) | | 0.05 | 1,201 (9.6%) | 172 (8.7%) | | 0.03 |
| Use of other lipid-lowering drugs; n (%) | 329 (8.9%) | 45 (7.5%) | 0.05 4 | 77 (16.2%) | 55 (12.8%) | 0.10 | 910 (15.6%) | 135 (14.3%) | | 0.04 | 1,716 (13.8% | 235 (11.9%) | | 0.06 |
| Use of statins; n (%) | 2,231 (60.6% | 374 (62.6%) | -0.04 2 | ,230 (75.9% | 342 (79.4%) | -0.08 | 4,610 (79.19 | 766 (81.4%) | | -0.06 | 9,071 (72.9% | 1,482 (75.3% | 6 | -0.05 |
| Use of thiazide; n (%) | 321 (8.7%) | 46 (7.7%) | 0.04 3 | 15 (10 7%) | 45 (10.4%) | 0.01 | 730 (12 5%) | 113 (12.0%) | | 0.02 | 1,366 (11.0% | 204 (10.4%) | | 0.02 |

# Table 1 Matched

| | | | | MATCHED | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Optum | | IIIATCHES | Marketscan | | | Medicare | | | Pooled | |
| Variable | Leuprolide | Degarelix | St. Diff | Leuprolide | Degarelix | St. Diff | Leuprolide | Degarelix | St. Diff | Leuprolide | Degarelix | St. Diff |
| Number of patients | 546 | 546 | | 415 | 415 | | 926 | 926 | | 1,887 | 1,887 | 7 |
| Year of Cohort Entry Date2008-2009: n (%) | | | | | | | | | | | | |
| 2008-2009; n (%)<br>2010; n (%) | 18 (3.3%) | 20 (3.7%) | -0.02 | 2 28 (6.7%) | 24 (5.8%) | 0.00 | 46 (5.0%) | 37 (4.0%) | 0.05 | 92 (4.9%) | 81 (4.3%) | 0.03 |
| 2011; n (%) | 26 (4.8%) | 23 (4.2%) | 0.02 | 3 42 (10.1%) | 45 (10.8%) | -0.02 | 2 53 (5.7%) | 49 (5.3%) | 0.03 | 121 (6.4%) | 117 (6.2%) | 0.03 |
| 2012; n (%) | 42 (7.7%) | 40 (7.3%) | | 2 44 (10.6%) | 50 (12.0%) | | 92 (9.9%) | 69 (7.5%) | | 178 (9.4%) | 159 (8.4%) | 0.04 |
| 2013; n (%) | 50 (9.2%) | 50 (9.2%) | 0.00 | | 56 (13.5%) | | 116 (12.5%) | 121 (13.1%) | -0.02 | 227 (12.0%) | 227 (12.0%) | 0.00 |
| 2014; n (%) | 39 (7.1%) | 35 (6.4%) | 0.03 | 42 (10.1%) | 46 (11.1%) | | 143 (15.4%) | 170 (18.4%) | | 224 (11.9%) | 251 (13.3%) | -0.04 |
| 2015; n (%) | 39 (7.1%) | 42 (7.7%) | | 2 58 (14.0%) | 60 (14.5%) | | 182 (19.7%) | 171 (18.5%) | | 279 (14.8%) | 273 (14.5%) | 0.01 |
| 2016; n (%) | 67 (12.3%) | 62 (11.4%) | | 63 (15.2%) | 63 (15.2%) | | 130 (14.0%) | 144 (15.6%) | | 260 (13.8%) | 269 (14.3%) | -0.01 |
| 2017; n (%) | 65 (11.9%)<br>72 (13.2%) | 74 (13.6%)<br>76 (13.9%) | -0.05 | 53 (12.8%) | 47 (11.3%)<br>24 (5.8%) | 0.05 | 164 (17.7%) | 165 (17.8%) | 0.00 | 282 (14.9%) | 286 (15.2%) | -0.01 |
| 2018; n (%)<br>2019; n (%) | 72 (13.2%)<br>89 (16.3%) | 91 (16.7%) | -0.02 | 2 24 (5.8%) | 24 (5.8%) | 0.00 | ***** | ***** | | | | + |
| 2019, ft (%) | 39 (7.1%) | 33 (6.0%) | 0.04 | 1 | | | | | | | | + |
| Age | 33 (7.1%) | 33 (0.0%) | 0.0- | 1 | | | | | | | | + |
| mean (sd) | 76.19 (6.92) | 76.04 (7.59) | 0.02 | 74.65 (9.34) | 74.49 (9.17) | 0.02 | 76.99 (6.56) | 77.02 (6.47) | 0.00 | 76.24 (6.74) | 76.18 (6.87) | 0.01 |
| median [IQR] | 77.00 [72.00, 81.00] | 76.00 [71.00, 82.00] | 0.14 | 75.00 [67.00, 82.00] | 75.00 [68.00, 82.00] | 0.00 | 76.00 [72.00, 82.00] | 77.00 [72.00, 82.00] | -0.15 | 76.07 (7.36) | 76.27 (7.46) | -0.03 |
| Region | | | | | | | | | | | | |
| 1 - Northeast; n (%) | 86 (15.8%) | 85 (15.6%) | | 94 (22.7%) | 92 (22.2%) | | 194 (21.0%) | 189 (20.4%) | | 374 (19.8%) | 366 (19.4%) | 0.01 |
| 2 - North Central; n (%) | 131 (24.0%) | 131 (24.0%) | | 145 (34.9%) | 144 (34.7%) | | 208 (22.5%) | 223 (24.1%) | | 484 (25.6%) | 498 (26.4%) | -0.02 |
| 3 - South; n (%)<br>4 - West; n (%) | 209 (38.3%)<br>120 (22.0%) | 205 (37.5%)<br>125 (22.9%) | 0.02 | 2 139 (33.5%)<br>2 37 (8.9%) | 130 (31.3%)<br>49 (11.8%) | | 373 (40.3%)<br>151 (16.3%) | 368 (39.7%)<br>146 (15.8%) | | 721 (38.2%)<br>308 (16.3%) | 703 (37.3%)<br>320 (17.0%) | -0.02 |
| 4 - West; n (%) | 120 (22.076) | 123 (22.376) | -0.02 | 3/ (0.370) | 42 (11.070) | -0.10 | 122 (10.5%) | 140 (13.0%) | 0.01 | 300 (10.370) | J2U (17.U%) | -0.02 |
| White; n (%) | 437 (80.0%) | 438 (80.2%) | -0.01 | il | | 1 | 796 (86.0%) | 803 (86.7%) | -0.02 | 1,233 (65.3%) | 1,241 (65.8%) | -0.01 |
| Asian; n (%) | 8 (1.5%) | 11 (2.0%) | -0.04 | | ***** | | N/A | N/A | N/A | N/A | N/A | N/A |
| Black; n (%) | 66 (12.1%) | 61 (11.2%) | 0.03 | | | | 93 (10.0%) | 85 (9.2%) | 0.03 | 159 (8.4%) | 146 (7.7%) | 0.03 |
| Hispanic; n (%) | 35 (6.4%) | 36 (6.6%) | -0.01 | | | | N/A | N/A | N/A | N/A | N/A | N/A |
| North American Native; n (%) | | | | | | | N/A | N/A | N/A | N/A | N/A | N/A |
| Other; n (%) | | | | | | - | 18 (1.9%) | 16 (1.7%) | 0.02 | 18 (1.9%) | 16 (1.7%) | 0.02 |
| Cardiovascular event prognosticators Acute or Old MI; n (%) | 204 (37.4%) | 212 (38.8%) | .n n: | 3 97 (23.4%) | 94 (22.7%) | 0.03 | 357 (38.6%) | 348 (37.6%) | 0.02 | 658 (34.9%) | 654 (34.7%) | 0.00 |
| Anxiety; n (%) | 32 (5.9%) | 33 (6.0%) | 0.00 | | 22 (5.3%) | | 60 (6.5%) | 57 (6.2%) | | 112 (5.9%) | 112 (5.9%) | 0.00 |
| Atrial Fibrillation; n (%) | 84 (15.4%) | 90 (16.5%) | | 8 62 (14.9%) | 70 (16.9%) | | 187 (20.2%) | 206 (22.2%) | | 333 (17.6%) | 366 (19.4%) | -0.05 |
| Coronary Atherosclerosis; n (%) | 436 (79.9%) | 432 (79.1%) | 0.02 | 305 (73.5%) | 302 (72.8%) | 0.02 | 764 (82.5%) | 762 (82.3%) | 0.01 | 1,505 (79.8%) | 1,496 (79.3%) | 0.01 |
| Coronary, Carotid, Illiac, Femoral, and Popliteal Revascularization (Angioplasty/Stent/CABG); n (%) | 30 (5.5%) | 43 (7.9%) | | 40 (9.6%) | 32 (7.7%) | | 63 (6.8%) | 70 (7.6%) | | 133 (7.0%) | 145 (7.7%) | -0.03 |
| Diabetes with Complications; n (%) | 181 (33.2%) | 186 (34.1%) | | 62 (14.9%) | 58 (14.0%) | | 745 (80.5%) | 724 (78.2%) | | 988 (52.4%) | 968 (51.3%) | 0.02 |
| Diabetes without Complications; n (%) | 98 (17.9%) | 116 (21.2%) | | 3 149 (35.9%) | 134 (32.3%) | | 340 (36.7%) | 351 (37.9%) | | 587 (31.1%) | 601 (31.8%) | -0.02 |
| DVT; n (%) | 24 (4.4%) | 23 (4.2%) | | 7 (1.7%) | 6 (1.4%)<br>28 (6.7%) | | 45 (4.9%) | 42 (4.5%)<br>135 (14.6%) | | 76 (4.0%) | 71 (3.8%) | 0.01 |
| Edema; n (%) Erectile dysfunction; n (%) | 60 (11.0%)<br>79 (14.5%) | 60 (11.0%)<br>77 (14.1%) | 0.00 | 30 (7.2%) | 42 (10.1%) | | 136 (14.7%) | 121 (13.1%) | 0.00 | 226 (12.0%)<br>239 (12.7%) | 223 (11.8%)<br>240 (12.7%) | 0.01 |
| Foot ulcer; n (%) | 12 (2.2%) | 18 (3.3%) | | 7 9 (2.2%) | 10 (2.4%) | | 48 (5.2%) | 48 (5.2%) | | 69 (3.7%) | 76 (4.0%) | -0.02 |
| Hyperlipidemia; n (%) | 459 (84.1%) | 467 (85.5%) | -0.04 | 300 (72.3%) | 290 (69.9%) | | 837 (90.4%) | 843 (91.0%) | | 1,596 (84.6%) | 1,600 (84.8%) | -0.01 |
| Hypertension; n (%) | 477 (87.4%) | 479 (87.7%) | -0.01 | 313 (75.4%) | 318 (76.6%) | -0.03 | 862 (93.1%) | 867 (93.6%) | | 1,652 (87.5%) | 1,664 (88.2%) | -0.02 |
| Intracranial or Retroperitoneal Hemorrhage; n (%) | 7 (1.3%) | 5 (0.9%) | | 4 (1.0%) | 3 (0.7%) | | 12 (1.3%) | 17 (1.8%) | | 23 (1.2%) | 25 (1.3%) | -0.01 |
| Ischemic Heart Disease; n (%) | 461 (84.4%) | 457 (83.7%) | | 325 (78.3%) | 319 (76.9%) | | 795 (85.9%) | 791 (85.4%) | | 1,581 (83.8%) | 1,567 (83.0%) | 0.02 |
| Ischemic Stroke; n (%) | 101 (18.5%) | 101 (18.5%) | | 77 (18.6%) | 76 (18.3%) | | 228 (24.6%) | 229 (24.7%) | 0.00 | 406 (21.5%) | 406 (21.5%) | 0.00 |
| Major Trauma; n (%) Obesity; n (%) | 21 (3.8%)<br>66 (12.1%) | 27 (4.9%)<br>59 (10.8%) | -0.09 | 5 22 (5.3%)<br>1 55 (13.3%) | 18 (4.3%)<br>45 (10.8%) | 0.05 | 65 (7.0%)<br>8 147 (15.9%) | 55 (5.9%)<br>159 (17.2%) | 0.04<br>-0.03 | 108 (5.7%)<br>268 (14.2%) | 100 (5.3%)<br>263 (13.9%) | 0.02 |
| Other Disorders of Thyroid Gland; n (%) | 12 (2.2%) | 16 (2.9%) | | 1 16 (3.9%) | 45 (10.8%)<br>13 (3.1%) | | 34 (3.7%) | 38 (4.1%) | | 62 (3.3%) | 67 (3.6%) | -0.02 |
| Overweight; n (%) | 38 (7.0%) | 40 (7.3%) | | 10 (2.4%) | 13 (3.1%) | | 41 (4.4%) | 42 (4.5%) | | 89 (4.7%) | 95 (5.0%) | -0.02 |
| PE: n (%) | 10 (1.8%) | 8 (1.5%) | | 2 (0.5%) | 2 (0.5%) | | N/A | N/A | N/A | N/A | N/A | N/A |
| Peripheral Vascular Disease; n (%) | 191 (35.0%) | 185 (33.9%) | 0.02 | 109 (26.3%) | 111 (26.7%) | -0.01 | 284 (30.7%) | 272 (29.4%) | 0.03 | 584 (30.9%) | 568 (30.1%) | 0.02 |
| Stable Angina; n (%) | 62 (11.4%) | 75 (13.7%) | | 7 38 (9.2%) | 34 (8.2%) | | 107 (11.6%) | 112 (12.1%) | | 207 (11.0%) | 221 (11.7%) | -0.02 |
| Systemic Embolism; n (%) | 9 (1.6%) | 8 (1.5%) | | 9 (2.2%) | 9 (2.2%) | | N/A | N/A | N/A | N/A | N/A | N/A |
| TIA; n (%) | 19 (3.5%) | 19 (3.5%) | 0.00 | 8 (1.9%) | 10 (2.4%) | -0.03 | 35 (3.8%) | 36 (3.9%) | -0.01 | 62 (3.3%) | 65 (3.4%) | -0.01 |
| General Health/Mortality Prognosticators Abnormal liver function; n (%) | 57 (10.4%) | 53 (9.7%) | 0.00 | 2 31 (7.5%) | 27 (6.5%) | 2.24 | 103 (11.1%) | 97 (10.5%) | 0.03 | 191 (10.1%) | 177 (9.4%) | 0.02 |
| Abnormal liver function; n (%) Alcohol Abuse/Dependence: n (%) | 19 (3.5%) | 53 (9.7%)<br>15 (2.7%) | | 5 5 (1.2%) | 27 (6.5%)<br>5 (1.2%) | | 18 (1.9%) | 97 (10.5%)<br>19 (2.1%) | | 191 (10.1%)<br>42 (2.2%) | 1// (9.4%)<br>39 (2.1%) | 0.02 |
| Anemias (Sickle-Cell, G6PD Deficiency, Nutrient Deficiency); n (%) | 129 (23.6%) | 141 (25.8%) | | 81 (19.5%) | 68 (16.4%) | 0.08 | 282 (30.5%) | 280 (30.2%) | | 492 (26.1%) | 489 (25.9%) | 0.00 |
| Asthma; n (%) | 23 (4.2%) | 21 (3.8%) | | 2 21 (5.1%) | 21 (5.1%) | | 60 (6.5%) | 58 (6.3%) | | 104 (5.5%) | 100 (5.3%) | 0.01 |
| COPD; n (%) | 127 (23.3%) | 125 (22.9%) | 0.03 | 84 (20.2%) | 74 (17.8%) | 0.06 | 236 (25.5%) | 221 (23.9%) | 0.04 | 447 (23.7%) | 420 (22.3%) | 0.03 |
| Delirium; n (%) | 15 (2.7%) | 14 (2.6%) | | 4 (1.0%) | 4 (1.0%) | | 34 (3.7%) | 34 (3.7%) | | 53 (2.8%) | 52 (2.8%) | 0.00 |
| Dementia; n (%) | 17 (3.1%) | 18 (3.3%) | | 11 (2.7%) | 9 (2.2%) | | 24 (2.6%) | 30 (3.2%) | | 52 (2.8%) | 57 (3.0%) | -0.01 |
| Depression; n (%) | 49 (9.0%) | 45 (8.2%) | 0.03 | 3 23 (5.5%) | 22 (5.3%) | | 72 (7.8%) | 76 (8.2%) | -0.01 | 144 (7.6%) | 143 (7.6%) | 0.00 |
| Falls; n (%) Fractures; n (%) | 31 (5.7%)<br>35 (6.4%) | 38 (7.0%)<br>29 (5.3%) | -0.05 | 5 10 (2.4%)<br>5 22 (5.3%) | 10 (2.4%)<br>21 (5.1%) | 0.00 | 60 (6.5%) | 71 (7.7%)<br>45 (4.9%) | -0.05 | 101 (5.4%)<br>101 (5.4%) | 119 (6.3%)<br>95 (5.0%) | -0.04<br>0.02 |
| HIV/AIDS; n (%) | 0 (0.0%) | 2 (0.4%) | -n no | 0 (0.0%) | 0 (0.0%) | N/A | N/A | 45 (4.9%)<br>N/A | N/A | N/A | N/A | N/A |
| Organ Transplant; n (%) | 1 (0.2%) | 3 (0.5%) | -0.05 | 4 (1.0%) | 4 (1.0%) | | N/A | N/A | N/A | N/A | N/A | N/A |
| Osteoporosis; n (%) | 29 (5.3%) | 23 (4.2%) | | 14 (3.4%) | 12 (2.9%) | | 48 (5.2%) | 54 (5.8%) | | 91 (4.8%) | 89 (4.7%) | 0.00 |
| Peptic Ulcer Disease; n (%) | 142 (26.0%) | 141 (25.8%) | | 73 (17.6%) | 72 (17.3%) | | 249 (26.9%) | 254 (27.4%) | | 464 (24.6%) | 467 (24.7%) | 0.00 |
| Pneumonia; n (%) | 19 (3.5%) | 15 (2.7%) | | 11 (2.7%) | 15 (3.6%) | | 18 (1.9%) | 19 (2.1%) | | 48 (2.5%) | 49 (2.6%) | -0.01 |
| Renal Failure; n (%) | 123 (22.5%) | 127 (23.3%) | -0.02 | | 56 (13.5%) | | 246 (26.6%) | 246 (26.6%) | | 425 (22.5%) | 429 (22.7%) | 0.00 |
| Renal Failure (CKD Stage 4 or higher); n (%) Sleep Apnea; n (%) | 17 (3.1%)<br>46 (8.4%) | 17 (3.1%)<br>52 (9.5%) | 0.00 | 10 (2.4%) | 12 (2.9%)<br>43 (10.4%) | | 47 (5.1%)<br>96 (10.4%) | 49 (5.3%)<br>106 (11.4%) | -0.01 | 74 (3.9%)<br>184 (9.8%) | 78 (4.1%)<br>201 (10.7%) | -0.01<br>-0.03 |
| Sleep Apnea; n (%) Sleep Disorder; n (%) | 46 (8.4%)<br>27 (4.9%) | 29 (5.3%) | | 2 26 (6.3%) | 43 (10.4%)<br>38 (9.2%) | | 96 (10.4%)<br>82 (8.9%) | 106 (11.4%) | | 184 (9.8%) | 201 (10.7%)<br>168 (8.9%) | -0.03 |
| Smoking: n (%) | 184 (33.7%) | 178 (32.6%) | | 2 73 (17.6%) | 66 (15.9%) | | 270 (29.2%) | 290 (31.3%) | | 527 (27.9%) | 534 (28.3%) | -0.00 |
| Frailty Score: Empirical Version 365 days (ICD-9 and ICD-10) v2 | ( | (32.070) | 3.02 | | (-3.370) | 0.0. | (23.270) | (32.3/9) | -0.03 | (-7.579) | | 3.01 |
| mean (sd) | 0.16 (0.05) | 0.16 (0.05) | 0.00 | 0.16 (0.05) | 0.16 (0.05) | 0.00 | 0.19 (0.06) | 0.19 (0.06) | 0.00 | 0.17 (0.05) | 0.17 (0.05) | 0.00 |
| median [IQR] | 0.15 [0.13, 0.19] | 0.16 [0.13, 0.19] | -0.20 | 0.15 [0.13, 0.18] | 0.15 [0.13, 0.19] | 0.00 | 0.18 [0.15, 0.22] | 0.18 [0.15, 0.22] | 0.00 | 0.16 (0.06) | 0.17 (0.06) | -0.17 |
| Healthcare utilization | | | | | | | | | | | | |
| Any hospitalization; n (%) | 109 (20.0%) | 133 (24.4%) | | 89 (21.4%) | 90 (21.7%) | -0.01 | 242 (26.1%) | 244 (26.3%) | | 440 (23.3%) | 467 (24.7%) | -0.03 |
| Bone mineral density; n (%) | 23 (4.2%) | 20 (3.7%) | 0.0 | 3 11 (2.7%) | 9 (2.2%) | | 41 (4.4%) | 41 (4.4%) | 0.00 | 75 (4.0%) | 70 (3.7%) | 0.02 |
| BUN tests; n (%) Cardiologist visit | 82 (15.0%) | 82 (15.0%) | 0.00 | 55 (13.3%) | 45 (10.8%) | 0.08 | 181 (19.5%) | 183 (19.8%) | -0.01 | 318 (16.9%) | 310 (16.4%) | 0.01 |
| O O | 203 (37.2%) | 189 (34.6%) | 0.0 | 181 (43.6%) | 187 (45.1%) | -n n | 200 (21.6%) | 194 (21.0%) | 0.01 | 584 (30.9%) | 570 (30.2%) | 0.02 |
| 1-2 | 160 (29.3%) | 164 (30.0%) | | 2 114 (27.5%) | 108 (26.0%) | | 336 (36.3%) | 320 (34.6%) | | 610 (32.3%) | 592 (31.4%) | 0.02 |
| 3-5 | 132 (24.2%) | 131 (24.0%) | | 75 (18.1%) | 75 (18.1%) | | 241 (26.0%) | 249 (26.9%) | | 448 (23.7%) | 455 (24.1%) | -0.03 |
| >=6 | 51 (9.3%) | 62 (11.4%) | | 45 (10.8%) | 45 (10.8%) | | 149 (16.1%) | 163 (17.6%) | | 245 (13.0%) | 270 (14.3%) | -0.04 |
| Colonoscopy; n (%) | 67 (12.3%) | 65 (11.9%) | 0.01 | 44 (10.6%) | 41 (9.9%) | | 91 (9.8%) | 108 (11.7%) | -0.06 | 202 (10.7%) | 214 (11.3%) | -0.02 |
| colonoscopy, ii (70) | | | | | | | | | | | | |
| Endocrinologist Visit; n (%) Fecal occult blood (FOB) test; n (%) | 17 (3.1%)<br>53 (9.7%) | 19 (3.5%)<br>47 (8.6%) | | 2 13 (3.1%)<br>1 16 (3.9%) | 15 (3.6%)<br>19 (4.6%) | | 70 (7.6%)<br>8 62 (6.7%) | 90 (9.7%)<br>64 (6.9%) | | 100 (5.3%)<br>131 (6.9%) | 124 (6.6%)<br>130 (6.9%) | -0.09 |

# Table 1 Matched

| Flu vaccine: n (%) | 222 (40.7%) | 204 (37.4%) | 0.07 84 (20.2%) | 79 (19.0%) | 0.02 | 599 (64.7%) | 605 (65.3%) | .0.0 | 905 (48.0%) | 888 (47.1%) | 0.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Glucose test strips; n (%) | 6 (1.1%) | 12 (2.2%) | -0.09 8 (1.9%) | 8 (1.9%) | | 59 (6.4%) | 63 (6.8%) | | 73 (3.9%) | 83 (4.4%) | -0.0 |
| Glucose tests; n (%) | 74 (13.6%) | 91 (16.7%) | -0.09 73 (17.6%) | 54 (13.0%) | | 268 (28.9%) | 271 (29.3%) | | 415 (22.0%) | 416 (22.0%) | 0.0 |
| HbA1c tests : n (%) | 246 (45.1%) | 249 (45.6%) | -0.01 101 (24.3%) | 92 (22.2%) | | 712 (76.9%) | 712 (76.9%) | | 1,059 (56.1%) | 1.053 (55.8%) | 0.0 |
| Imaging/Diagnostics Used in Prostate Cancer | 240 (43.176) | 249 (43.0%) | -0.01 101 (24.3%) | 32 (22.270) | 0.03 | 712 (70.370) | 712 (70.376) | 0.00 | 1,033 (30.170) | 1,055 (55.6%) | 0.0 |
| n o nagriostics osed in Frostate Cancer | 177 (32.4%) | 181 (33.2%) | -0.02 128 (30.8%) | 132 (31.8%) | -0.02 | 332 (35.9%) | 348 (37.6%) | -0.0 | 637 (33.8%) | 661 (35.0%) | -0.0 |
| 1.2 | 304 (55.7%) | 296 (54.2%) | 0.03 209 (50.4%) | 208 (50.1%) | | 449 (48.5%) | 433 (46.8%) | | 962 (51.0%) | 937 (49.7%) | 0.0 |
| 20 | 65 (11.9%) | 69 (12.6%) | -0.02 78 (18.8%) | 75 (18.1%) | | 145 (15.7%) | 145 (15.7%) | | 288 (15.3%) | 289 (15.3%) | 0.0 |
| Internal Medicine/Family Medicine Visits; n (%) | 512 (93.8%) | 521 (95.4%) | -0.07 368 (88.7%) | 364 (87.7%) | | 827 (89.3%) | 824 (89.0%) | | 1,707 (90.5%) | 1,709 (90.6%) | 0.0 |
| Lipid tests; n (%) | 407 (74.5%) | 402 (73.6%) | 0.02 151 (36.4%) | 146 (35.2%) | | 770 (83.2%) | 775 (83.7%) | | 1,328 (70.4%) | 1,323 (70.1%) | 0.0 |
| Microalbuminuria tests; n (%) | 129 (23.6%) | 138 (25.3%) | -0.04 70 (16.9%) | 66 (15.9%) | | 423 (45.7%) | 419 (45.2%) | | 622 (33.0%) | 623 (33.0%) | 0.0 |
| | 129 (23.6%) | 136 (23.3%) | -0.04 70 (16.9%) | 00 (13.9%) | 0.03 | 423 (43.7%) | 419 (43.270) | 0.0. | 022 (33.0%) | 623 (33.0%) | 0.0 |
| Number of different/distinct medication prescriptionsmean (sd) | 8.05 (5.80) | 8.22 (6.03) | -0.03 10.77 (5.60) | 10.45 (5.00) | 0.06 | 11.62 (4.86) | 11.67 (4.91) | 0.0 | 10.40 (4.84) | 10.40 (4.79) | 0.0 |
| median [IQR] | 8.00 [4.00, 12.00] | 8.00 [4.00, 12.00] | 0.00 10.00 [7.00, 14.00] | 10.00 [7.00, 13.00] | | 11.00 [8.00, 15.00] | 11.00 [8.00, 15.00] | | 9.91 (5.31) | 9.91 (5.28) | 0.0 |
| Office Visits (outpatient setting only) | 8.00 [4.00, 12.00] | 8.00 [4.00, 12.00] | 0.00 10.00 [7.00, 14.00] | 10.00 [7.00, 13.00] | 0.00 | 11.00 [8.00, 15.00] | 11.00 [8.00, 15.00] | 0.00 | 9.91 (5.51) | 9.91 (5.28) | 0.0 |
| | 12.19 (6.15) | 12.35 (6.28) | -0.03 13.06 (6.91) | 12.48 (6.36) | 0.00 | 13.78 (6.87) | 14.30 (6.98) | 0.01 | 13.16 (5.92) | 13.34 (5.86) | -0.0 |
| mean (sd) | 11.00 [8.00, 15.00] | 11.00 [8.00, 15.00] | 0.00 12.00 [8.00, 16.00] | 11.00 [8.00, 16.00] | | 13.00 [9.00, 17.00] | 13.00 [9.00, 18.00] | | 12.20 (6.68) | 11.98 (6.65) | 0.0 |
| median [IQR] Oncology Specialist Visit | 11.00 [8.00, 15.00] | 11.00 [8.00, 15.00] | 0.00 12.00 [8.00, 16.00] | 11.00 [8.00, 16.00] | 0.15 | 13.00 [9.00, 17.00] | 13.00 [9.00, 18.00] | 0.00 | 12.20 (6.68) | 11.98 (6.65) | 0.0 |
| Oncology Specialist Visit | 370 (67.8%) | 370 (67.8%) | 0.00 3.00 (00.30/) | 375 (90.4%) | 0.05 | F.C.F. (C.4. 00/.) | F 4 C (F 0 00/) | 2.2 | 1.303 (69.1%) | 1,291 (68,4%) | 0.0 |
| | | | 0.00 368 (88.7%) | | | 565 (61.0%) | 546 (59.0%) | | | | |
| 1-5 | 73 (13.4%) | 72 (13.2%) | 0.01 18 (4.3%) | 16 (3.9%) | | 166 (17.9%) | 181 (19.5%) | | 257 (13.6%) | 269 (14.3%) | -0.0 |
| >=6 | 103 (18.9%) | 104 (19.0%) | 0.00 29 (7.0%) | 24 (5.8%) | | 195 (21.1%) | 199 (21.5%) | | 327 (17.3%) | 327 (17.3%) | 0.0 |
| Pneumonia vaccine; n (%) | 174 (31.9%) | 174 (31.9%) | 0.00 45 (10.8%) | 48 (11.6%) | -0.03 | 257 (27.8%) | 275 (29.7%) | -0.0 | 476 (25.2%) | 497 (26.3%) | -0.0 |
| Prostate cancer prognosticators | (2.20) | - // | | L., | 1 | | | | L.,. | | |
| Radiation Therapies Used in Prostate Cancer; n (%) | 3 (0.5%) | 1 (0.2%) | 0.05 1 (0.2%) | 0 (0.0%) | 0.06 | N/A | N/A | N/A | N/A | N/A | N/A |
| PSA Test | | | | | | | | | | | |
| mean (sd) | 2.38 (1.80) | 2.41 (1.75) | -0.02 0.94 (1.45) | 1.01 (1.53) | | 2.33 (1.40) | 2.40 (1.42) | | 2.04 (1.40) | 2.10 (1.41) | 0.0 |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.25] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | | 1.56 (1.54) | 1.56 (1.55) | 0.0 |
| Prostatectomy; n (%) | 14 (2.6%) | 17 (3.1%) | -0.03 16 (3.9%) | 11 (2.7%) | -0.24 | 22 (2.4%) | 21 (2.3%) | -0.2 | 52 (2.8%) | 49 (2.6%) | 0.0 |
| Prostate exam for DRE | | | | | | | | | | | |
| mean (sd) | 1.27 (3.29) | 1.17 (2.84) | 0.03 0.33 (1.34) | 0.30 (1.42) | 0.02 | 0.45 (0.90) | 0.42 (0.82) | 0.0 | 0.66 (1.94) | 0.61 (1.72) | 0.0 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.98) | 0.00 (1.76) | 0.0 |
| Prostate Cancer Comorbidity Index (PCCI) | | | | | | | | | | | |
| mean (sd) | 36.39 (6.41) | 36.50 (6.31) | -0.02 34.75 (5.72) | 34.42 (5.19) | | 37.00 (6.38) | 36.99 (6.21) | 0.00 | 36.33 (5.55) | 36.28 (5.35) | 0.0 |
| median [IQR] | 35.00 [32.00, 40.00] | 35.00 [32.00, 40.00] | 0.00 34.00 [30.00, 38.00] | 34.00 [30.00, 37.00] | 0.00 | 36.00 [32.00, 41.00] | 36.00 [33.00, 41.00] | 0.00 | 35.27 (6.25) | 35.27 (6.03) | 0.0 |
| Medications | | | | | | | | | | | |
| ACE inhibitors; n (%) | 179 (32.8%) | 178 (32.6%) | 0.00 162 (39.0%) | 173 (41.7%) | -0.06 | 446 (48.2%) | 453 (48.9%) | -0.0: | 787 (41.7%) | 804 (42.6%) | -0.0 |
| Anti-arrhythmics; n (%) | 9 (1.6%) | 11 (2.0%) | -0.03 7 (1.7%) | 5 (1.2%) | 0.04 | 11 (1.2%) | 19 (2.1%) | -0.0 | 27 (1.4%) | 35 (1.9%) | -0.0 |
| Anti-diabetic Drugs; n (%) | 116 (21.2%) | 114 (20.9%) | 0.01 114 (27.5%) | 111 (26.7%) | | 582 (62.9%) | 574 (62.0%) | | 812 (43.0%) | 799 (42.3%) | 0.0 |
| Chemotherapies Used in Prostate Cancer; n (%) | 3 (0.5%) | 1 (0.2%) | 0.05 1 (0.2%) | 0 (0.0%) | 0.06 | N/A | N/A | N/A | N/A | N/A | N/A |
| Metformin; n (%) | 73 (13.4%) | 77 (14.1%) | -0.02 76 (18.3%) | 62 (14.9%) | 0.09 | 320 (34.6%) | 341 (36.8%) | -0.0 | 469 (24.9%) | 480 (25.4%) | -0.0 |
| Use of anticonvulsants: n (%) | 46 (8.4%) | 49 (9.0%) | -0.02 44 (10.6%) | 41 (9.9%) | 0.02 | 128 (13.8%) | 135 (14.6%) | -0.0 | 218 (11.6%) | 225 (11.9%) | -0.0 |
| Use of antidepressants; n (%) | 67 (12.3%) | 64 (11.7%) | 0.02 46 (11.1%) | 53 (12.8%) | -0.05 | 144 (15.6%) | 142 (15.3%) | 0.0 | 257 (13.6%) | 259 (13.7%) | 0.0 |
| Use of Antiparkinsonian Meds; n (%) | 10 (1.8%) | 10 (1.8%) | 0.00 6 (1.4%) | 7 (1.7%) | | 20 (2.2%) | 18 (1.9%) | | 36 (1.9%) | 35 (1.9%) | 0.0 |
| Use of antiplatelet agents; n (%) | 143 (26.2%) | 142 (26.0%) | 0.00 164 (39.5%) | 153 (36.9%) | | 358 (38.7%) | 348 (37.6%) | | 665 (35.2%) | 643 (34.1%) | 0.0 |
| Use of antipsychotics: n (%) | 6 (1.1%) | 6 (1.1%) | 0.00 4 (1.0%) | 7 (1.7%) | -0.06 | | | N/A | N/A | N/A | N/A |
| Use of anxiolytics/hypnotics; n (%) | 24 (4.4%) | 23 (4.2%) | 0.01 22 (5.3%) | 24 (5.8%) | | 57 (6.2%) | 62 (6.7%) | | 103 (5.5%) | 109 (5.8%) | -0.0 |
| Use of ARBs; n (%) | 81 (14.8%) | 87 (15.9%) | -0.03 90 (21.7%) | 86 (20.7%) | | 248 (26.8%) | 228 (24.6%) | | 419 (22.2%) | 401 (21.3%) | 0.0 |
| Use of Benzos; n (%) | 51 (9.3%) | 54 (9.9%) | -0.02 48 (11.6%) | 44 (10.6%) | | 98 (10.6%) | 103 (11.1%) | | 197 (10.4%) | 201 (10.7%) | -0.0 |
| Use of beta blockers; n (%) | 273 (50.0%) | 278 (50.9%) | -0.02 268 (64.6%) | 276 (66.5%) | | 668 (72.1%) | 675 (72.9%) | | 1,209 (64.1%) | 1,229 (65.1%) | -0.0 |
| Use of bisphosphonate; n (%) | 12 (2.2%) | 9 (1.6%) | 0.04 11 (2.7%) | 5 (1.2%) | | 18 (1.9%) | 18 (1.9%) | | 41 (2.2%) | 32 (1.7%) | 0.0 |
| Use of calcium channel blockers; n (%) | 144 (26.4%) | 144 (26.4%) | 0.00 110 (26.5%) | 108 (26.0%) | | 288 (31.1%) | 291 (31.4%) | | . 542 (28.7%) | 543 (28.8%) | 0.0 |
| Use of COPD/asthma meds; n (%) | 75 (13.7%) | 78 (14.3%) | -0.02 93 (22.4%) | 82 (19.8%) | | 172 (18.6%) | 163 (17.6%) | | 340 (18.0%) | 323 (17.1%) | 0.0 |
| Use of Dementia Meds; n (%) | 6 (1.1%) | 8 (1.5%) | -0.04 11 (2.7%) | 8 (1.9%) | | 20 (2.2%) | 19 (2.1%) | | 37 (2.0%) | 35 (1.9%) | -0.0 |
| Use of digoxin; n (%) | 9 (1.6%) | 10 (1.8%) | -0.02 11 (2.7%) | 12 (2.9%) | | 31 (3.3%) | 43 (4.6%) | | 51 (2.7%) | 65 (3.4%) | |
| Use of heparin and other low-molecular weight heparins; n (%) | 4 (0.7%) | 6 (1.1%) | -0.04 9 (2.2%) | 6 (1.4%) | | 26 (2.8%) | 25 (2.7%) | | 39 (2.1%) | 37 (2.0%) | 0.0 |
| Use of Insulin; n (%) | 23 (4.2%) | 28 (5.1%) | -0.04 30 (7.2%) | 32 (7.7%) | | 174 (18.8%) | 184 (19.9%) | | 227 (12.0%) | 244 (12.9%) | -0.0 |
| Use of Lithium; n (%) | 1 (0.2%) | 0 (0.0%) | 0.06 0 (0.0%) | 0 (0.0%) | | N/A | | N/A | N/A | N/A | N/A |
| Use of Loop Diuretics; n (%) | 45 (8.2%) | 52 (9.5%) | -0.05 51 (12.3%) | 58 (14.0%) | | 186 (20.1%) | 195 (21.1%) | | 282 (14.9%) | 305 (16.2%) | -0.0 |
| Use of nitrates; n (%) | 74 (13.6%) | 69 (12.6%) | 0.03 74 (17.8%) | 77 (18.6%) | | 198 (21.4%) | 201 (21.7%) | | 346 (18.3%) | 347 (18.4%) | 0.0 |
| Use of NSAIDs; n (%) | 71 (13.0%) | 69 (12.6%) | 0.01 62 (14.9%) | 57 (13.7%) | | 141 (15.2%) | 128 (13.8%) | | 274 (14.5%) | 254 (13.5%) | 0.0 |
| Use of opioids; n (%) | 169 (31.0%) | 159 (29.1%) | 0.04 158 (38.1%) | 162 (39.0%) | | 376 (40.6%) | 361 (39.0%) | | 703 (37.3%) | 682 (36.1%) | 0.0 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, Apixaban, Warfarin); n (%) | 46 (8.4%) | 46 (8.4%) | 0.00 51 (12.3%) | 51 (12.3%) | | 138 (14.9%) | 147 (15.9%) | | 235 (12.5%) | 244 (12.9%) | -0.0 |
| | 126 (23.1%) | 124 (22.7%) | 0.01 110 (26.5%) | 100 (24.1%) | | 277 (29.9%) | 246 (26.6%) | | 513 (27.2%) | 470 (24.9%) | 0.0 |
| Use of oral corticosteroids; n (%) | | | 0.06 4 (1.0%) | 3 (0.7%) | 0.03 | N/A | N/A | N/A | N/A | N/A | N/A |
| Use of other antiplatelet agents; n (%) | 8 (1.5%) | 5 (0.9%) | | | | | | | | | |
| Use of other antiplatelet agents; n (%) | 8 (1.5%)<br>16 (2.9%) | 5 (0.9%)<br>16 (2.9%) | 0.06 4 (1.0%) | 21 (5.1%) | | 48 (5.2%) | 51 (5.5%) | -0.0 | 93 (4.9%) | 88 (4.7%) | 0.0 |
| Use of other antiplatelet agents; n (%) | | | | | 0.08 | 48 (5.2%)<br>96 (10.4%) | 51 (5.5%)<br>90 (9.7%) | | 93 (4.9%) | 88 (4.7%)<br>168 (8.9%) | 0.0 |
| Use of other antiplatelet agents; n (%) Use of other diuretics; n (%) | 16 (2.9%) | 16 (2.9%) | 0.00 29 (7.0%) | 21 (5.1%) | 0.08<br>-0.03 | | | 0.02 | | | |
| Use of other antiplatelet agents; n (%) Use of other diuretics; n (%) Use of other diuretics; n (%) Use of other hypertension drugs; n (%) | 16 (2.9%)<br>44 (8.1%) | 16 (2.9%)<br>47 (8.6%) | 0.00 29 (7.0%)<br>-0.02 28 (6.7%) | 21 (5.1%)<br>31 (7.5%) | 0.08<br>-0.03<br>-0.05 | 96 (10.4%) | 90 (9.7%) | 0.03<br>-0.03 | 168 (8.9%) | 168 (8.9%) | 0.0 |